CLINICAL TRIAL: NCT00533897
Title: A Phase IIIb, Multi-Center, Randomized, Withdrawal Study to Evaluate the Immunogenicity and Safety of Subcutaneous Administered Abatacept in Adults With Active Rheumatoid Arthritis
Brief Title: Phase IIIB Subcutaneous Missed Dose Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-167
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2011-06-03 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abatacept (Experimental)
  Interventions: Drug: Abatacept
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abatacept — Solution in pre-filled syringes, Subcutaneously, 125 mg, Weekly, (Short Term (3 periods - 12 weeks each; Long Term)
  Other Names: Orencia; BMS-188667
  Arms: Abatacept
Drug: Placebo — Solution in pre-filled syringes, Subcutaneously, 0 mg, Weekly, Period II 12 weeks (Short Term)
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether subcutaneous abatacept administered to patients with rheumatoid arthritis is associated with increased immunogenicity or increased safety events upon withdrawal and reintroduction.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Rheumatoid Arthritis
* Disease Activity Score (DAS)28-C-Reactive Protein (CRP) score ≥ 3.2 and ≤5.1
* On background methotrexate at least 3 months (≥10mg weekly)
* Must be able to self injection or allow a care giver to do it for them
* Discontinue all Biologics and Disease-Modifying Anti-rheumatic Drugs (DMARDs) except for methotrexate

Exclusion Criteria:

* Participants who had prior exposure to abatacept or CTLA-4 Ig
* Received treatment with rituximab.
* Participants who have received treatment with leflunomide within 1 year of screening
* Participants who have received treatment with immunoadsorption columns (such as Prosorba columns), mycophenolate mofetil (Cellcept®), cyclosporine A or other calcineurin inhibitors, or D-Penicillamine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- United States (13):
  - Wallace Rheumatic Study Center, Los Angeles, California
  - New England Research Associates, Llc, Trumbull, Connecticut
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Diagnostic Rheumatology And Research,Pc, Indianapolis, Indiana
  - Klein And Associates, M.D., Pa, Cumberland, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - St. Paul Rheumatology, P.A., Eagan, Minnesota
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - East Penn Rheumatology Associates, Bethlehem, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Center For Assessment And Research Of Erie, Erie, Pennsylvania
  - Columbia Arthritis Center, Columbia, South Carolina
  - Mountain State Clinical Research, Clarksburg, West Virginia
- Argentina (4):
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Santa Fe, Santa Fe Province
- Local Institution, Trois-Rivières, Quebec, Canada
- Mexico (4):
  - Local Institution, León, Guanajuato
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Metepec, State of Mexico
  - Local Institution, Mérida, Yucatán
- South Africa (5):
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Muckleneuk, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Berea, KwaZulu-Natal
  - Local Institution, Panorama, Western Cape

REFERENCES:
- [Derived] Kaine J, Gladstein G, Strusberg I, Robles M, Louw I, Gujrathi S, Pappu R, Delaet I, Pans M, Ludivico C. Evaluation of abatacept administered subcutaneously in adults with active rheumatoid arthritis: impact of withdrawal and reintroduction on immunogenicity, efficacy and safety (phase Iiib ALLOW study). Ann Rheum Dis. 2012 Jan;71(1):38-44. doi: 10.1136/annrheumdis-2011-200344. Epub 2011 Sep 13. PMID 21917824

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Rheumatoid Arthritis (American College of Rheumatology Class I, II or III) were enrolled. Study initiated November 2007. Short Term (ST) results and some long term extension (LTE) results up to a database lock in 2010 were released earlier. Study concluded February 2014. Final LTE results are now included.
Pre-assignment Details: 270 participants enrolled; 167 were treated in the Short Term (ST) study. 103 were not treated (10 withdrew consent, 2 lost to follow-up, 91 no longer met study criteria). ST study included 3 Periods: Lead-In (LI), Doubleblind Withdrawal (DBW), and Reintroduction (RI).150 participants entered the LTE study.
Groups:
- Abatacept (ABA) [Lead-In (LI)]: On Day 1 of the 12 week Lead-In (LI), participants received a single intravenous (IV) ABA dose based on participant weight (<60 kg=500 mg, 60-100 kg=750 mg, >100 kg=1 g). Following, participants received weekly subcutaneous (SC) of open-label ABA (fixed dose of 125 mg) through Day 78.
- Abatacept (ABA) Double-blind Withdrawal (DBW): After receiving ABA in the LI, participants received double blind ABA SC injections (fixed dose of 125 mg) starting on Day 85 and weekly for 12 weeks.
- Placebo (PLA) Double Blind Withdrawal (DBW): After receiving ABA in the LI Period, participants received double blind Placebo SC injections starting on Day 85 and weekly for 12 weeks.
- ABA With IV PLA Loading Dose in Re-introduction (RI) Period: After receiving ABA in LI Period, and ABA in DBW Period, participants received a single blinded placebo IV dose on Day 169 and continued with weekly SC injections of open-label ABA for 12 weeks (fixed dose of 125 mg) in the RI Period.
- PLA Switched to ABA With ABA IV Loading Dose in RI Period: After receiving ABA in LI period, and PLA in the DBW Period, participants were randomized to receive a single weight-titered ABA IV loading dose (<60 kg=500 mg, 60-100 kg=750 mg, >100 kg=1 g) followed by weekly open-label SC ABA injections (fixed dose of 125 mg) in the RI Period.
- PLA Switched to ABA With PLA IV Loading Dose in RI Period: After receiving ABA in the Lead-In, and PLA in the DBW Period, participants were randomized to receive a single Placebo IV loading dose on Day 169 followed by weekly open-label SC ABA injections (fixed dose of 125 mg) in the RI Period.
- Long Term Extension Abatacept for LI Period Non-responders: Participants received Abatacept SC injections (fixed dose of 125 mg) during Lead-in (LI) Period 1 for 12 weeks. If after 12 weeks the participant was a non-responder (unable to achieve Disease Activity Score 28 (DAS28-CRP) decrease by ≥ 0.6 from Day 1), they directly entered the Long Term Extension (LTE) receiving open label Abatacept SC injections (125 mg) starting on Day 85 and weekly for 12 weeks (ie, participants did not enter DBW or RI periods). If clinical response was achieved, participant continued in LTE until SC administration of Abatacept was approved by the respective country and commercially available or until sponsor elected to terminate the study.
- Long Term Extension (LTE) Abatacept for Short Term Completers: Participant's who successfully completed the Short Term of the study, could enter the LTE on Day 253 and receive weekly open-label SC abatacept (125 mg) in the LTE until SC administration of ABA was approved by the respective country and commercially available or until the sponsor elected to terminate the study. Participants who completed the ST study (Completers) had received ABA during LI Period 1, entered DBW Period 2 (ABA or PLA), and in RI Period 3 continued/switched to ABA (with either ABA or PLA IV loading dose, as appropriate).
Period: Lead-in (LI) Period 1
Arm/Group | Abatacept (ABA) [Lead-In (LI)] | Abatacept (ABA) Double-blind Withdrawal (DBW) | Placebo (PLA) Double Blind Withdrawal (DBW) | ABA With IV PLA Loading Dose in Re-introduction (RI) Period | PLA Switched to ABA With ABA IV Loading Dose in RI Period | PLA Switched to ABA With PLA IV Loading Dose in RI Period | Long Term Extension Abatacept for LI Period Non-responders | Long Term Extension (LTE) Abatacept for Short Term Completers
Started | 167 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 157 (37 participants entered the LTE directly and did not enter the DBW Period nor receive DBW treatment.) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Withdrew Consent | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Administrative Reason By Sponsor | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Missed 2 Consecutive Doses of Study Drug | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double-blind Withdrawal (DBW) Period 2
Arm/Group | Abatacept (ABA) [Lead-In (LI)] | Abatacept (ABA) Double-blind Withdrawal (DBW) | Placebo (PLA) Double Blind Withdrawal (DBW) | ABA With IV PLA Loading Dose in Re-introduction (RI) Period | PLA Switched to ABA With ABA IV Loading Dose in RI Period | PLA Switched to ABA With PLA IV Loading Dose in RI Period | Long Term Extension Abatacept for LI Period Non-responders | Long Term Extension (LTE) Abatacept for Short Term Completers
Started | 0 | 40 | 80 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 39 (One participant discontinued the DBW Period due to Lack of Efficacy to enter the RI Period early) | 77 (Two participants discontinued the DBW Period due to Lack of Efficacy to enter the RI Period early) | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Poor/Non-Compliance | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Re-introduction (RI) Period 3
Arm/Group | Abatacept (ABA) [Lead-In (LI)] | Abatacept (ABA) Double-blind Withdrawal (DBW) | Placebo (PLA) Double Blind Withdrawal (DBW) | ABA With IV PLA Loading Dose in Re-introduction (RI) Period | PLA Switched to ABA With ABA IV Loading Dose in RI Period | PLA Switched to ABA With PLA IV Loading Dose in RI Period | Long Term Extension Abatacept for LI Period Non-responders | Long Term Extension (LTE) Abatacept for Short Term Completers
Started | 0 | 0 | 0 | 40 (1 participant discontinued the DBW Period due to Lack of Efficacy to enter RI Period early) | 35 (1 participant discontinued the DBW Period due to Lack of Efficacy to enter RI Period early) | 44 (1 participant discontinued the DBW Period due to Lack of Efficacy to enter RI Period early) | 0 | 0
Completed | 0 | 0 | 0 | 40 | 35 | 42 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Participant Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — No Longer Meets Study Criteria | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Long Term Extension (LTE)
Arm/Group | Abatacept (ABA) [Lead-In (LI)] | Abatacept (ABA) Double-blind Withdrawal (DBW) | Placebo (PLA) Double Blind Withdrawal (DBW) | ABA With IV PLA Loading Dose in Re-introduction (RI) Period | PLA Switched to ABA With ABA IV Loading Dose in RI Period | PLA Switched to ABA With PLA IV Loading Dose in RI Period | Long Term Extension Abatacept for LI Period Non-responders | Long Term Extension (LTE) Abatacept for Short Term Completers
Started | 0 | 0 | 0 | 0 | 0 | 0 | 37 (37 non-responders in Lead-In entered the LTE directly and didn't participate in DBW or RI Periods.) | 113 (117 completed RI but 4 did not enter LTE: 1 lack of efficacy and 3 had their site closed.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 24 (Participant continued until SC ABA was available in respective country or Sponsor ended study.) | 88 (Participant continued until SC ABA was available in respective country or Sponsor ended study.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 25
Not completed — Participant Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3
Not completed — Poor/Non-compliance | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6

BASELINE CHARACTERISTICS:
Population: All Period 1 Non-responders and Period 2 participants who received at least one dose of abatacept during the study were summarized.
Groups:
- Period 1 Non-Responders: Participants received abatacept (ABA) intravenous (IV) loading dose and subcutaneous (SC) injections (fixed dose of 125 mg abatacept) on Day 1 followed by weekly SC injections of ABA up to Day 85 during the Lead-in Period (Period 1). Period 1 non-responders skipped Periods 2 and 3 and entered the long term extension (LTE).
- Abatacept Received in Period 2: Participants received ABA IV loading dose and SC injections (fixed dose of 125 mg abatacept) on Day 1 followed by weekly SC injections of ABA up to Day 85 during the Lead-in Period (Period 1). Period 1 responders continued into Period 2 and were randomized to ABA (Day 85-169).
- Placebo Received in Period 2: Participants received ABA IV loading dose and SC injections (fixed dose of 125 mg abatacept) on Day 1 followed by weekly SC injections of ABA up to Day 85 during the Lead-in Period (Period 1). Period 1 responders continued into Period 2 and were randomized to Placebo (Day 85-169).
- Total: Total of all reporting groups
Arm/Group | Period 1 Non-Responders | Abatacept Received in Period 2 | Placebo Received in Period 2 | Total
Number analyzed (Participants) | 37 | 40 | 80 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (12.7) | 48.9 (14.2) | 49.1 (12.8) | 49.8 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 34 | 67 | 131
  Male | 7 | 6 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Withdrawal (DBW) Period; Percentage of Participants With Positive Anti-Abatacept or Anti-Cytotoxic T-Lymphocyte Antigen 4 (CTLA4) Antibody Responses by Enzyme-Linked Immunosorbent Assay (ELISA) at Day 169
Description: Serum samples from all treated adult participants with active rheumatoid arthritis (RA) were screened for the presence of drug-specific antibodies using an enzyme-linked immunosorbent assay (ELISA). Immunogenicity was defined as the presence of a positive anti-abatacept or anti-CTLA4 antibody.
Time Frame: Day 169
Population: Participants treated in the DBW Period with at least 1 immunogenicity result (ELISA) during DBW Period. N=Number of Participants Analyzed, n=number of participants with data for that time point
Measure: Number; unit: percentage of participants
Groups:
- Abatacept in DBW Period: Participants received Abatacept (ABA) SC injections (fixed dose of 125 mg) starting on Day 85 and weekly for 12 weeks
- Placebo in DBW Period: Participants received placebo (PLA) SC injections starting on Day 85 and weekly for 12 weeks.
Arm/Group | Abatacept in DBW Period | Placebo in DBW Period
Number analyzed (Participants) | 40 | 80
percentage of participants
  Anti-abatacept (n=37, n=71) | 0 | 1.4
  Anti-CTLA4-T (n=38, n=73) | 0 | 8.2
  Total (n=38, n=73) | 0 | 9.6
Statistical Analysis 1: Comparison: Abatacept in DBW Period vs Placebo in DBW Period; A continuity corrected Chi-square test was used to compare percentage of positive antibody responses of SC placebo vs. SC abatacept (Period II treatment groups) on Day 169. P-value was evaluated at 0.05 significance level (2-sided). 95% confidence interval (CI) for difference (SC PLA - SC ABA) between ABA and PLA in the immunogenicity rates was also calculated. Point estimates of the immunogenicity rates within the two Period II treatment group and the corresponding 95% CIs were also provided; Test type: Superiority or Other; p = 0.119, Chi-squared, Corrected — There was no adjustment made for multiple comparisons; estimate of difference = 9.59, 95% CI 2-sided [0.83 to 18.34]

2. Secondary Outcome: RI Period; Percentage of Participants With Positive Anti-Abatacept or Anti-CTLA4 Antibody Responses by ELISA at Day 253, by DBW Period Placebo Group
Description: Serum samples from Abatacept-treated adult participants with active RA were screened for the presence of drug-specific antibodies using ELISA. Immunogenicity was defined as the presence of a positive anti-abatacept or anti-CTLA4 antibody.
Time Frame: Day 253 (short term)
Population: Participants treated with Placebo in DBW period who were treated in RI period and had at least 1 immunogenicity result (ELISA) during RI period. N=Number of Participants Analyzed, n=number of participants with data for that time point
Measure: Number; unit: percentage of participants
Groups:
- PLA Switched to ABA With ABA IV Loading Dose in RI Period: On Day 169, participants were randomized to receive a single ABA IV loading dose based on participant weight (<60 kg=500 mg, 60-100 kg=750 mg, >100 kg=1 g) and weekly open-label SC ABA injections (fixed dose of 125 mg) were re-introduced in the RI Period.
- PLA Switched to ABA With PLA IV Loading Dose in RI Period: On Day 169, participants were randomized to receive a single PLA IV loading dose and weekly open-label SC ABA injections (fixed dose of 125 mg) were re-introduced in the RI Period.
Arm/Group | PLA Switched to ABA With ABA IV Loading Dose in RI Period | PLA Switched to ABA With PLA IV Loading Dose in RI Period
Number analyzed (Participants) | 35 | 44
percentage of participants
  Anti-abatacept (n=32, n=41) | 0 | 0
  Anti-CTLA4-T (n=32, n=41) | 0 | 4.9
  Total (n=32, n=41) | 0 | 4.9
Statistical Analysis 1: Comparison: PLA Switched to ABA With ABA IV Loading Dose in RI Period vs PLA Switched to ABA With PLA IV Loading Dose in RI Period; Immunogenicity rates of the Period II treatment groups on Day 253 were analyzed similarly as on Day 169. However, no statistical test was carried out and no p-value was provided. Provided were: point estimates of the immunogenicity rates within the Period II treatment groups and corresponding 95% CIs, and point estimate for the difference in immunogenicity rates between these groups and corresponding 95% CI. There was no adjustment made for multiple comparisons; Test type: Superiority or Other; Estimate of Difference = 4.88, 95% CI 2-sided [-4.50 to 14.25]

3. Secondary Outcome: Lead-in (LI) Period; Percentage of Participants With Positive Anti-Abatacept or Anti-CTLA4 Antibody Responses by ELISA Over Time
Description: as for outcome 2
Time Frame: For on-treatment visits: Day 1-Day 85, includes ≤21 Days after last dose or up to 1st dose of DBW Period. For follow-up post visits for participants who discontinued drug in LI: Day 22 after last dose of drug to Day 85 after last dose of drug
Population: All participants treated in LI Period who had at least 1 immunogenicity result (ELISA) during LI period. N=Number of Participants Analyzed, n=number of participants with data for that time point
Measure: Number; unit: percentage of participants
Groups:
- Abatacept in Lead-In Period: On Day 1, participants received a single intravenous (IV) Abatacept (ABA) dose based on participant weight (<60 kg=500 mg, 60-100 kg=750 mg, >100 kg=1 g). Following, participants received weekly subcutaneous (SC) of open-label ABA (fixed dose of 125 mg) through Day 78.
Arm/Group | Abatacept in Lead-In Period
Number analyzed (Participants) | 167
percentage of participants
  Overall on TRT visits: anti-ABA (n=162) | 1.2
  Overall on TRT visits: anti-CTLA4 (n=165) | 0
  Overall on TRT visits: Total (n=165) | 1.2
  Overall post visits: anti-ABA (n=3) | 0
  Overall post visits: anti-CTLA4 (n=3) | 0
  Overall post visits: Total (n=3) | 0
  Overall anti-ABA (n=162) | 1.2
  Overall anti-CTLA4 (n=165) | 0
  Overall Total (n=165) | 1.2

4. Secondary Outcome: LI Period; Percentage of Participants With Positive Anti-Abatacept or Anti-CTLA4 Antibody Responses by Electrochemiluminescence (ECL) Over Time
Description: ECL screened sera for drug-specific antibodies; immunocompetition was used to identify specific anti-Abatacept reactivity. Cytotoxic leukocyte antigen 4 (CTLA4) and Possibly Immunoglobulin (Ig) Category=reactivity against extracellular domain of human CTLA4, constant regions of human IgG1, or both (CTLA4Ig; Abatacept molecule). Ig and/or Junction (JNC) Category=reactivity against constant regions and/or hinge region of human IgG1. Drug-induced seropositivity was defined as a post-baseline titer higher than Baseline, or any post-baseline positivity if Baseline value was missing or negative.
Time Frame: as for outcome 3
Population: All participants treated in Period 1 (Lead-in Period). N=Number of Participants Analyzed, n=number of participants with data for that time point
Measure: Number; unit: percentage of participants
Groups:
- Abatacept in Lead-In Period: On Day 1, participants received a single intravenous (IV) ABA dose based on participant weight (<60 kg=500 mg, 60-100 kg=750 mg, >100 kg=1 g). Following, participants received weekly subcutaneous (SC) of open-label ABA (fixed dose of 125 mg) through Day 78.
Arm/Group | Abatacept in Lead-In Period
Number analyzed (Participants) | 167
percentage of participants
  Overall onTRT visits CTLA4 and Possibly Ig, n=165 | 1.2
  Overall onTRT visits Ig and/or JNC region, n=165 | 0
  Overall onTRT visits Total, n=165 | 1.2
  Overall post visits CTLA4 and possibly Ig, n=3 | 0
  Overall post visits Ig and/or JNC region, n=3 | 0
  Overall post visits: Total, n=3 | 0
  Overall CTLA4 and possibly Ig, n=165 | 1.2
  Overall Ig and/or JNC region, n=165 | 0
  Overall Total (n=165) | 1.2

5. Secondary Outcome: DBW Period; Percentage of Participants With Positive Anti-Abatacept or Anti-CTLA4 Antibody Responses by ELISA Over Time
Description: Serum samples from Abatacept-treated adult participants with active RA were screened for the presence of drug-specific antibodies using ELISA. Immunogenicity was defined as the presence of a positive anti-abatacept or anti-CTLA4 antibody. Samples were obtained during treatment (TRT) visits.
Time Frame: Days 86-169, includes ≤21 Days after last dose or up to 1st dose of RI Period
Population: All participants treated in DBW period with at least 1 immunogenicity result (ELISA) during DBW period. N=Number of Participants Analyzed, n=number of participants with data for that time point.
Measure: Number; unit: percentage of participants
Groups:
- Abatacept in DBW Period: Participants received ABA SC injections (fixed dose of 125 mg) starting on Day 85 and weekly for 12 weeks.
- Placebo in DBW Period: Participants received PLA SC injections starting on Day 85 and weekly for 12 weeks.
Arm/Group | Abatacept in DBW Period | Placebo in DBW Period
Number analyzed (Participants) | 40 | 80
percentage of participants
  Overall on TRT visits: anti-ABA, n=39,78 | 0 | 1.3
  Overall on TRT visits anti-CTLA4, n=40,80 | 0 | 7.5
  Overall on TRT visits: Total, n=40,80 | 0 | 8.8

6. Primary Outcome: Re-introduction (RI) Period; Percentage of Participants With Positive Anti-Abatacept or Anti-CTLA4 Antibody Responses by ELISA at Day 253, by DBW Period Groups
Description: as for outcome 2
Time Frame: Day 253 (short term)
Population: Participants treated in RI period with at least 1 immunogenicity result (ELISA) during RI period. N=Number of Participants Analyzed, n=number of participants with data for that time point.
Measure: Number; unit: percentage of participants
Groups:
- ABA in DBW Period: Participants received ABA SC injections (fixed dose of 125 mg) starting on Day 85 and weekly for 12 weeks
Arm/Group | ABA in DBW Period | Placebo in DBW Period
Number analyzed (Participants) | 40 | 79
percentage of participants
  Anti-abatacept (n=38, n=73) | 0 | 0
  Anti-CTLA4-T (n=38, n=73) | 2.6 | 2.7
  Total (n=38, n=73) | 2.6 | 2.7
Statistical Analysis 1: Comparison: ABA in DBW Period vs Placebo in DBW Period; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Estimate of Difference = 0.11, 95% CI 2-sided [-8.21 to 8.43]

7. Secondary Outcome: DBW Period; Percentage of Participants With Positive Anti-Abatacept or Anti-CTLA4 Antibody Responses by ELISA at Post Visits
Description: as for outcome 2
Time Frame: Day 22 after last dose of drug to Day 85 after last dose of drug
Population: These data were not summarized since there were no participants at any post visits.
Groups:
- PLA in DBW Period: Participants received PLA SC injections starting on Day 85 and weekly for 12 weeks.
Arm/Group | ABA in DBW Period | PLA in DBW Period
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: DBW Period; Percentage of Participants With Positive Anti-Abatacept or Anti-CTLA4 Antibody Responses by ECL Over Time
Description: as for outcome 4
Time Frame: Days 86-169, includes ≤21 Days after last dose or up to 1st dose of RI Period
Population: All participants treated in DBW period with at least 1 immunogenicity result (ECL) during DBW period. N=Number of Participants Analyzed, n=number of participants with data for that time point
Measure: Number; unit: percentage of participants
Arm/Group | ABA in DBW Period | PLA in DBW Period
Number analyzed (Participants) | 40 | 80
percentage of participants
  Overall onTRT visits CTLA4 and Possibly Ig,n=40,80 | 0 | 6.3
  Overall onTRT visits Ig and/or JNC region, n=40,80 | 0 | 3.8
  Overall on TRT visits: Total Abs, n=40,80 | 0 | 10.0

9. Secondary Outcome: DBW Period; Percentage of Participants With Positive Anti-Abatacept or Anti-CTLA4 Antibody Responses by ECL At Post Visits
Description: as for outcome 4
Time Frame: Day 22 after last dose of drug to Day 85 after last dose of drug
Population: These data were not summarized since there were no participants at any post visits
Arm/Group | ABA in DBW Period | PLA in DBW Period
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: RI Period; Percentage of Participants With Positive Anti-Abatacept or Anti-CTLA4 Antibody Responses by ELISA Over Time by DBW Treatment Group
Description: as for outcome 2
Time Frame: For on-treatment visits: Days 170-253, includes ≤21 Days after last dose or up to 1st dose of LTE Period. For follow-up post visits for participants who discontinued drug in RI: Day 22 after last dose of drug to Day 85 after last dose of drug
Population: All participants treated in RI period with at least 1 immunogenicity result (ELISA) during RI period N=Number of Participants Analyzed, n=number of participants with data for that time point.
Measure: Number; unit: percentage of participants
Groups:
- ABA [DBW]: Participants received ABA SC injections (fixed dose of 125 mg) starting on Day 85 and weekly for 12 weeks.
- PLA [DBW]: Participants received PLA SC injections starting on Day 85 and weekly for 12 weeks.
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 79
percentage of participants
  Overall onTRT visits: anti-ABA, n=39,77 | 2.6 | 1.3
  Overall onTRT visits anti-CTLA4, n=40,78 | 5.0 | 3.8
  Overall onTRT visits: Total, n=40,78 | 7.5 | 5.1
  Overall post visits: anti-ABA, n=1,4 | 0 | 0
  Overall post visits: anti-CTLA4, n=1,4 | 0 | 25.0
  Overall post visits: Total, n=1,4 | 0 | 25.0

11. Secondary Outcome: RI Period; Percentage of Participants With Positive Anti-Abatacept or Anti-CTLA4 Antibody Responses by ECL Over Time by DBW Treatment Group
Description: as for outcome 4
Time Frame: as for outcome 10
Population: All participants treated in RI period with at least 1 immunogenicity result (ECL) during RI period N=Number of Participants Analyzed, n=number of participants with data for that time point
Measure: Number; unit: percentage of participants
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 79
percentage of participants
  Overall onTRT visits CTLA4 and Possibly Ig,n=40,78 | 0 | 0
  Overall onTRT visits Ig and/or JNC region, n=40,78 | 0 | 0
  Overall onTRT visits: Total, n=40,78 | 0 | 0
  Overall post visits: CTLA4 and possibly Ig, n=1,4 | 100.0 | 25.0
  Overall post visits: Ig and/or JNC region, n=1,4 | 0 | 0
  Overall post visits: Total, n=1,4 | 100.0 | 25.0

12. Secondary Outcome: Short Term (ST); Percentage of Participants With Positive Anti-Abatacept or Anti-CTLA4 ELISA Antibody Responses by DBW Treatment Groups
Description: Serum samples from Abatacept-treated adult participants with active rheumatoid arthritis (RA) were screened for the presence of drug-specific antibodies using ELISA. Immunogenicity was defined as the presence of a positive anti-abatacept or anti-CTLA4 antibody. ST was defined as the LI Period, the DBW Period, and the RI Period (Days 1-253).
Time Frame: For on-TRT visits: Days 1-253 (ST). For follow-up post visits for participants who discontinued drug in the ST: Day 22 after last dose of ST drug to Day 85 after last dose of ST drug
Population: All participants treated in DBW period with at least 1 immunogenicity result (ELISA) during the Short Term. N=Number of Participants Analyzed, n=number of participants with data for that time point.
Measure: Number; unit: percentage of participants
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 80
percentage of participants
  Overall study onTRT visits: anti-ABA, n=39,78 | 7.7 | 1.3
  Overall study onTRT visits anti-CTLA4, n=40,80 | 5.0 | 8.8
  Overall study onTRT visits: Total, n=40,80 | 12.5 | 10.0
  Overall study post visits: anti-ABA, n=1, 4 | 0 | 0
  Overall study post visits: anti-CTLA4, n=1, 4 | 0 | 25.0
  Overall study post visits: Total, n=1, 4 | 0 | 25.0
  Overall study anti-ABA, n=39, 78 | 7.7 | 1.3
  Overall study anti-CTLA4, n=40, 80 | 5.0 | 8.8
  Overall study Total, n=40,80 | 12.5 | 10.0

13. Secondary Outcome: Short Term: Percentage of Participants With Positive Anti-Abatacept or Anti-CTLA4 ECL Antibody Responses by DBW Treatment Groups
Description: as for outcome 4
Time Frame: as for outcome 12
Population: All participants treated in DBW period with at least 1 immunogenicity result (ECL) during the Short Term. N=Number of Participants Analyzed, n=number of participants with data for that time point.
Measure: Number; unit: percentage of Participants
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 80
percentage of Participants
  Overall onTRT visits CTLA and possibly Ig,n=40,80 | 0 | 7.5
  Overall onTRT visits Ig and/or JNC region,n=40,80 | 0 | 3.8
  Overall study onTRT visits: Total, n=40,80 | 0 | 10.0
  Overall post visits CTLA4 and possibly Ig,n=1,4 | 100.0 | 25.0
  Overall post visits: Ig and/or JNC region, n=1,4 | 0 | 0
  Overall study post visits: Total, n=1, 4 | 100.0 | 25.0
  Overall study CTLA4 and possibly Ig,n=40,80 | 2.5 | 8.8
  Overall study Ig and/or JNC region, n=40, 80 | 0 | 3.8
  Overall study Total, n=40,80 | 2.5 | 11.3

14. Secondary Outcome: Short Term: Mean Change in Disease Activity Score (DAS) 28 (Using C-Reactive Protein [CRP]) From Baseline Over Time by DBW Treatment Groups
Description: The DAS28 is a continuous disease measure composite of 4 variables: the number of tender joints out of 28 joints, the number of swollen joints out of 28 joints, the level of the serum reactant protein CRP, and participant global assessment of disease activity measure on a visual analogue scale. DAS28 has numeric thresholds defining high disease activity (> 5.1), low disease activity (≤ 3.2) and remission (< 2.6). Clinically meaningful improvement= decrease in DAS28 score of ≥1.2 from baseline.
Time Frame: Days 1 (Baseline),15, 29, 57, 78, 85, 113, 141, 169, 197, 225, and 253 (short term)
Population: Intent To Treat Analysis Population (DBW Period, Participants randomized in DBW period who received at least 1 dose of study medication in DBW period). N=Number of Participants Analyzed, n=number of participants with data for that time point and at baseline.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 80
units on a scale
  Day 15, n=38, n=75 | -0.64 (0.10) | -0.87 (0.08)
  Day 29, n=40, n=80 | -1.07 (0.14) | -1.10 (0.09)
  Day 57, n=40. n=79 | -1.39 (0.14) | -1.62 (0.11)
  Day 78, n=33, n=76 | -1.76 (0.12) | -1.89 (0.10)
  Day 85, n=40, n=78 | -1.97 (0.11) | -1.88 (0.11)
  Day 113, n=39, n=80 | -1.78 (0.18) | -1.69 (0.12)
  Day 141, n=38, n=76 | -1.81 (0.17) | -1.54 (0.14)
  Day 169, n=38, n=75 | -2.03 (0.18) | -1.49 (0.14)
  Day 197, n=40, n=79 | -2.14 (0.16) | -1.92 (0.13)
  Day 225, n=39, n=77 | -2.20 (0.17) | -2.04 (0.13)
  Day 253, n=39, n=74 | -2.22 (0.14) | -2.32 (0.12)

15. Secondary Outcome: Short Term: Percentage of Participants Achieving Clinically Meaningful Improvement (CMI) in DAS 28 (CRP), Low Disease Activity (LDAS), or Clinical Remission Over Time by DBW Treatment Groups
Description: DAS28 is a continuous disease measure composite of 4 variables: the number of tender joints out of 28 joints, the number of swollen joints out of 28 joints, the level of the serum reactant protein CRP, and participant global assessment of disease activity measure on a visual analogue scale. DAS28 has numeric thresholds defining high disease activity (> 5.1), low disease activity (≤ 3.2) and remission (< 2.6). Clinically meaningful improvement= decrease in DAS28 score of ≥1.2 from baseline.
Time Frame: Days 85, 169, and 253 (short term)
Population: Intent To Treat Analysis Population (DBW Period, Participants randomized in DBW period who received at least 1 dose of study medication in DBW period). N=Number of Participants Analyzed, n=number of participants with data for that time point and, when relevant, at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 80
percentage of participants
  Day 85 CMI , n=40, n=78 | 80 | 76.9
  Day 85 LDAS, n=40, n=78 | 67.5 | 62.8
  Day 85 Clinical Remission, n=40, n=78 | 35.0 | 37.2
  Day 169 CMI , n=38, n=75 | 78.9 | 57.3
  Day 169 LDAS, n=38, n=75 | 68.4 | 54.7
  Day 169 Clinical Remission, n=38, n=75 | 47.4 | 28.0
  Day 253 CMI , n=39, n=74 | 87.2 | 89.2
  Day 253 LDAS, n=39, n=74 | 69.2 | 79.7
  Day 253 Clinical Remission, n=39, n=74 | 51.3 | 63.5

16. Secondary Outcome: Short Term; Mean Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) From Baseline Over Time by DBW Treatment Groups
Description: The disability section of the full HAQ includes 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. The questions are evaluated on a 4-point scale: 0=without any difficulty, 1= with some difficulty, 2= with much difficulty, and 3= unable to do. Higher scores= greater dysfunction. A disability index was calculated by summing the worst scores in each domain and dividing by the number of domains answered. Clinically meaningful HAQ response=an improvement of at least 0.3 units from baseline in HAQ disability Index.
Time Frame: Days 1 (Baseline),15, 29, 57, 78, 85, 113, 141, 169, 197, 225, and 253 (short term)
Population: as for outcome 14
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo (PLA) [DBW]: Participants received PLA SC injections starting on Day 85 and weekly for 12 weeks.
Arm/Group | ABA [DBW] | Placebo (PLA) [DBW]
Number analyzed (Participants) | 40 | 80
units on a scale
  Day 15, n=40, n=77 | -0.31 (0.06) | -0.30 (0.04)
  Day 29, n=40, n=80 | -0.46 (0.05) | -0.35 (0.04)
  Day 57, n=40, n=79 | -0.58 (0.09) | -0.51 (0.06)
  Day 78, n=33, n=77 | -0.68 (0.10) | -0.59 (0.07)
  Day 85, n=40, n=79 | -0.74 (0.09) | -0.63 (0.07)
  Day 113, n=40, n=80 | -0.69 (0.08) | -0.61 (0.06)
  Day 141, n=39, n=78 | -0.68 (0.10) | -0.52 (0.07)
  Day 169, n=38, n=76 | -0.72 (0.11) | -0.50 (0.07)
  Day 197, n=40, n=79 | -0.76 (0.09) | -0.66 (0.06)
  Day 225, n=40, n=77 | -0.82 (0.10) | -0.70 (0.06)
  Day 253, n=39, n=74 | -0.86 (0.09) | -0.72 (0.06)

17. Secondary Outcome: Short Term; Percentage of Participants With HAQ-DI Response Over Time by DBW Treatment Groups
Description: as for outcome 16
Time Frame: Days 1 (Baseline),15, 29, 57, 78, 85, 113, 141, 169, 197, 225, and 253 (short term)
Population: as for outcome 14
Measure: Number; unit: percentage of Participants
Groups:
- ABA [DB]: Participants received ABA SC injections (fixed dose of 125 mg) starting on Day 85 and weekly for 12 weeks
- PLA [DB]: Participants received PLA SC injections starting on Day 85 and weekly for 12 weeks.
Arm/Group | ABA [DB] | PLA [DB]
Number analyzed (Participants) | 40 | 80
percentage of Participants
  Day 15, n=40, n=77 | 47.5 | 42.9
  Day 29, n=40, n=80 | 62.5 | 52.5
  Day 57, n=40, n=79 | 67.5 | 62.0
  Day 78, n=33, n=77 | 66.7 | 67.5
  Day 85, n=40, n=79 | 80.0 | 69.6
  Day 113, n=40, n=80 | 75.0 | 67.5
  Day 141, n=39, n=78 | 69.2 | 62.8
  Day 169, n=38, n=76 | 71.1 | 56.6
  Day 197, n=40, n=79 | 75.0 | 74.7
  Day 225, n=40, n=77 | 80.0 | 76.6
  Day 253, n=39, n=74 | 84.6 | 74.3

18. Secondary Outcome: LI; Mean Change in DAS 28 (CRP) From Baseline Over Time
Description: as for outcome 15
Time Frame: Days 1 (Baseline), 15, 29, 57, 78, 85
Population: Participants who received at least 1 dose of study medication during LI period. N=Number of Participants Analyzed, n=number of participants with data for that time point and at baseline.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- ABA [LI]: On Day 1, participants received a single intravenous (IV) ABA dose based on participant weight (<60 kg=500 mg, 60-100 kg=750 mg, >100 kg=1 g). Following, participants received weekly subcutaneous (SC) of open-label ABA (fixed dose of 125 mg) through Day 78.
Arm/Group | ABA [LI]
Number analyzed (Participants) | 167
units on a scale
  Day 15, n=150 | -0.72 (0.06)
  Day 29, n=165 | -1.00 (0.07)
  Day 57, n=164 | -1.35 (0.08)
  Day 78, n=143 | -1.39 (0.10)
  Day 85, n=161 | -1.53 (0.10)

19. Secondary Outcome: LI; Percentage of Participants With Clinically Meaningful Improvement in DAS (CRP) Over Time
Description: as for outcome 15
Time Frame: Days 15, 29, 57, 78, 85
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | ABA [LI]
Number analyzed (Participants) | 167
percentage of participants
  Day 15, n=150 | 26.0
  Day 29, n=165 | 40.6
  Day 57, n=164 | 56.1
  Day 78, n=143 | 59.4
  Day 85, n=161 | 64.6

20. Secondary Outcome: DBW Period; Mean Change in DAS 28 (CRP) From DBW Period Baseline (Day 85) Over Time
Description: as for outcome 15
Time Frame: Days 85 (Period 2 Baseline), 113, 141, and 169
Population: Intent To Treat Analysis Population (DBW Period, Participants randomized in DBW period who received at least 1 dose of study medication in DBW period). N=Number of Participants Analyzed, n=number of participants with data for that time point and at DBW period baseline.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 80
units on a scale
  Day 113, n=39, n=76 | 0.19 (0.18) | 0.16 (0.11)
  Day 141 , n=38, n=73 | 0.14 (0.17) | 0.35 (0.15)
  Day 169, n=38, n=72 | -0.06 (0.19) | 0.40 (0.14)

21. Secondary Outcome: DBW Period; Percentage of Participants With Rheumatoid Arthritis (RA) Flare Over Time
Description: A participant had an RA flare if at least 2 of the following criteria were met:
  * Doubling of tender and swollen joint count from Day 78
  * Increase in DAS28-CRP score ≥ 1.2 from Day 78
  * Prematurely discontinued from Double-blind Withdrawal Period (Period 2) and continued to Re-introduction Period (Period 3)
Time Frame: Days 85, 113, 141, and 169
Population: Intent To Treat Analysis Population (DBW Period, Participants randomized in DBW period who received at least 1 dose of study medication in DBW period). N=Number of Participants Analyzed, n=number of participants with data for that time point.
Measure: Number; unit: percentage of participants
Arm/Group | ABA [DB] | PLA [DB]
Number analyzed (Participants) | 40 | 80
percentage of participants
  Day 85, n=31, n=66 | 0 | 1.5
  Day 113, n=33, n=77 | 9.1 | 2.6
  Day 141, n=32, n=73 | 6.3 | 6.8
  Day 169, n=33, n=74 | 6.1 | 9.5

22. Secondary Outcome: RI Period; Mean Change in DAS 28 (CRP) From RI Period Baseline (Day 169) Over Time
Description: as for outcome 15
Time Frame: Days 169 (Period III Baseline), 197, 225, and 253
Population: Participants who received at least 1 dose of study medication during RI period. N=Number of Participants Analyzed, n=number of participants with data for that time point and at RI period baseline.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- ABA With IV PLA Loading Dose [RI]: Participants received a single placebo IV dose on Day 169, and continued weekly SC injections of open-label ABA for 12 weeks (fixed dose of 125 mg).
- PLA Switched to ABA With ABA IV Loading Dose [RI]: Participants were randomized to receive a single ABA IV loading dose based on participant weight (<60 kg=500 mg, 60-100 kg=750 mg, >100 kg=1 g) and weekly open-label SC ABA injections (fixed dose of 125 mg) were re-introduced.
- PLA Switched to ABA With PLA IV Loading Dose [RI]: Participants were randomized to receive a single PLA IV loading dose and weekly open-label SC ABA injections (fixed dose of 125 mg) were re-introduced.
Arm/Group | ABA With IV PLA Loading Dose [RI] | PLA Switched to ABA With ABA IV Loading Dose [RI] | PLA Switched to ABA With PLA IV Loading Dose [RI]
Number analyzed (Participants) | 40 | 35 | 44
units on a scale
  Day 197, n=39, n=33, n=44 | -0.26 (0.17) | -0.56 (0.17) | -0.50 (0.16)
  Day 225, n=38, n=33, n=42 | -0.31 (0.20) | -0.59 (0.18) | -0.66 (0.17)
  Day 253, n=38, n=30, n=42 | -0.23 (0.16) | -0.93 (0.20) | -0.89 (0.17)

23. Secondary Outcome: LI; Number of Participants With Deaths, Serious Adverse Events (SAEs), SAEs Leading to Discontinuation, Adverse Events (AEs), Related AEs, or AEs Leading to Discontinuation
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event.
Time Frame: From Day 1 through Day 85, up to 56 days post last dose in Lead-in Period or up to first dose in next period, whichever occurred earlier
Population: Participants who received at least 1 dose of study medication during LI period
Measure: Number; unit: participants
Arm/Group | ABA [LI]
Number analyzed (Participants) | 167
participants
  Deaths | 1
  SAEs | 3
  Related SAEs | 0
  SAEs Leading to Discontinuation | 1
  AEs | 82
  Related AEs | 29
  AEs Leading to Discontinuation | 1

24. Secondary Outcome: LI Period; Number of Participants With AEs of Special Interest
Description: AEs of special interest are those AEs that may be associated with the use of immunomodulatory drugs, including all infections and opportunistic infections; autoimmune disorders; malignancies; acute infusional AEs (pre-specified AEs occurring within 1 hour of start of infusion), peri-infusional AEs (pre-specified AEs occurring within 24 hours of the start of infusion),local injection site reaction (pre-specified AEs occurring at the site of SC injection)and systemic injection site reactions (pre-specified systemic AEs such as hypersensitivity reactions occurring within 24 hours of SC injection)
Time Frame: as for outcome 23
Population: Participants who received at least 1 dose of study medication during LI period
Measure: Number; unit: participants
Arm/Group | ABA [LI]
Number analyzed (Participants) | 167
participants
  Infections and infestations | 42
  Malignancies | 0
  Autoimmune events (prespecified) | 0
  Acute infusional events (prespecified) | 1
  Peri-infusional events (prespecified) | 2
  Local injection site reactions (prespecified) | 2
  Systemic injection reactions (prespecified) | 9

25. Secondary Outcome: LI; Number of Participants With Hematology Values Meeting the Marked Abnormality (MA) Criteria
Description: Upper Normal Limit (ULN), Lower Normal Limit (LLN), Baseline (BL). Marked abnormality criteria are: Hemoglobin (HGB): >3 g/dL decrease from BL; Hematocrit: <0.75 * BL; Erythrocytes: <0.75 * BL; Platelets (PLT): <0.67 * LLN/>1.5 * ULN, or if BL < LLN then use <0.5 * BL and <100,000 mm^3; Leukocytes: <0.75 * LLN/ >1.25 * ULN, or if BL<LLN then use <0.8 * BL or >ULN, or if BL>ULN then use >1.2 * BL or <LLN; neutrophils+bands: <1.0 * 10^3 cells/ microliter (uL); eosinophils: >0.750 * 10^3 cells/uL; basophils: > 400 mm^3; monocytes: >2000 mm^3; lymphocytes: <0.750 * 10^3 cells/uL/ >7.50 * 10^3 cells/uL.
Time Frame: as for outcome 23
Population: Participants who received at least 1 dose of study medication during LI period.
Measure: Number; unit: participants
Arm/Group | ABA [LI]
Number analyzed (Participants) | 167
participants
  Low HGB | 0
  Low hematocrit | 0
  Low erythrocytes | 1
  Low PLT | 1
  High PLT | 0
  Low leukocytes | 3
  High leukocytes | 4
  Low neutrophils+bands | 0
  High eosinophils | 1
  High basophils | 0
  High monocytes | 0
  Low lymphocytes | 7
  High lymphocytes | 0

26. Secondary Outcome: LI; Number of Participants With Liver and Kidney Function Values Meeting the Marked Abnormality Criteria
Description: Marked abnormality criteria: Alkaline phosphatase (ALP): >2* ULN, or if BL>ULN then use >3* BL; aspartate aminotransferase (AST): >3* ULN, or if BL>ULN then use >4* BL; alanine aminotransferase (ALT): >3* ULN, or if BL>ULN then use >4* BL; G-Glutamyl transferase (GGT): >2* ULN, or if BL>ULN then use >3* BL; Bilirubin: >2* ULN, or if BL>ULN then use >4* BL; blood urea nitrogen (BUN): >2* BL; creatinine: >1.5* BL
Time Frame: as for outcome 23
Population: Participants who received at least 1 dose of study medication during LI period.
Measure: Number; unit: participants
Arm/Group | ABA [LI]
Number analyzed (Participants) | 167
participants
  High ALP | 0
  High AST | 1
  High ALT | 2
  High GGT | 0
  High bilirubin | 0
  High BUN | 1
  High creatinine | 3

27. Secondary Outcome: LI; Number of Participants With Electrolyte Values Meeting the Marked Abnormality Criteria
Description: Marked abnormality criteria: Sodium (Na): <0.95*LLN/ >1.05*ULN, or if BL<LLN then use <0.95* BL or >ULN, or if BL>ULN then use>1.05* BL or <LLN; potassium (K): <0.9* LLN/>1.1*ULN, or if BL<LLN then use <0.9* BL or >ULN, or if BL>ULN then use>1.1* BL or <LLN; (Cl): <0.9* LLN/>1.1* ULN, or if BL<LLN then use <0.9* BL or >ULN, or if BL>ULN then use>1.1* BL or <LLN; calcium (Ca): <0.8* LLN/>1.2* ULN, or if BL<LLN then use <0.75* BL or >ULN, or if BL>ULN then use>1.25* BL or <LLN; phosphorous (P): <0.75* LLN/ >1.25* ULN, or if BL<LLN then use 0.67* BL or >ULN, or if BL>ULN then use>1.33* BL or <LLN
Time Frame: as for outcome 23
Population: Participants who received at least 1 dose of study medication during LI period.
Measure: Number; unit: participants
Arm/Group | ABA [LI]
Number analyzed (Participants) | 167
participants
  Low Na | 0
  High Na | 0
  Low K | 0
  High K | 0
  Low Cl | 0
  High Cl | 0
  Low Ca | 0
  High Ca | 0
  Low P | 1
  High P | 1

28. Secondary Outcome: LI; Number of Participants With Other Chemistry and Urinalysis Values Meeting the Marked Abnormality Criteria
Description: MA criteria: serum glucose (Glu): <65 mg/dL/>220 mg/dL;fasting serum Glu: <0.8* LLN/>1.5*upper limits of normal (ULN),or if BL< lower limits of normal (LLN) then use 0.8*BL or > upper limits of normal (ULN),or if BL>ULN then use >2.0*BL or <LLN;total protein: <0.9*LLN/>1.1*ULN,or if BL<LLN then use <0.9*BL or >ULN,or if BL>UNL then use >1.1*BL or <LLN; albumin: <0.9*LLN,or if BL<LLN then use <0.75 BL;uric acid: >1.5*ULN,or if BL>ULN then use >2*BL. Urinalysis: Urine protein,urine Glu,urine blood,leukocyte esterase,Red Blood Cells (RBCs), White Blood Cells (WBCs):Use ≥2 when BL value missing or when pre-dose=0 or 0.5; use ≥3 when pre-dose=1, use ≥4 when pre-dose=2 or 3
Time Frame: as for outcome 23
Population: Participants who received at least 1 dose of study medication during LI period. N=Number of Participants Analyzed. n (when indicated)= number of participants with data available during LI period.
Measure: Number; unit: participants
Arm/Group | ABA [LI]
Number analyzed (Participants) | 167
participants
  Low Glu (n=167) | 9
  High Glu (n=167) | 4
  Low fasting Glu (n=92) | 3
  High fasting glucose (n=92) | 0
  Low protein (n=167) | 1
  High protein (n=167) | 1
  Low Albumin (n=167) | 0
  High uric acid (n=167) | 0
  High urine protein (n=167) | 3
  High urine Glu (n=167) | 3
  High urine blood (n=167) | 17
  High leukocyte esterase (n=46) | 9
  High urine RBC (n=44) | 7
  High urine WBC (n=63) | 26

29. Secondary Outcome: LI Period; Mean Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure was taken in participants while seated and measured in millimeters of mercury (mmHg). Pressures were assessed at screening, at baseline on Day 1 prior to infusion of IV abatacept, at 30 and 60 minutes after IV infusion of abatacept on Day 1, and at all office visits prior to SC injection of abatacept. Vital signs were also assessed 7 days after the last injection of abatacept for participants who were withdrawn prematurely.
Time Frame: Days 1, 15, 29, 57, 78, and 85
Population: Participants who received at least 1 dose of study medication during LI period. N=Number of Participants Analyzed. n (when indicated)= number of participants with data available at that time point during the LI period.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ABA [LI]
Number analyzed (Participants) | 167
mmHg
  Day 1 SBP before infusion (n=160) | 125.0 (18.42)
  Day 15 SBP before injection (n=156) | 122.3 (14.55)
  Day 29 SBP before injection (n=161) | 122.0 (14.02)
  Day 57 SBP before injection (n=157) | 121.4 (14.87)
  Day 78 SBP before injection (n=157) | 120.3 (14.38)
  Day 85 SBP before injection (n=159) | 122.0 (15.19)
  Day 1 DBP before infusion (n=160) | 76.0 (10.88)
  Day 15 DBP before injection (n=156) | 75.8 (9.63)
  Day 29 DBP before injection (n=161) | 76.1 (9.43)
  Day 57 DBP before injection (n=157) | 75.7 (9.82)
  Day 78 DBP before injection (n=157) | 75.4 (10.29)
  Day 85 DBP before injection (n=159) | 75.2 (9.45)

30. Secondary Outcome: LI Period; Mean Heart Rate (HR)
Description: Heart rate was taken in participants while seated and measured in beats per minute (bpm). Heart rate was assessed at screening, at baseline on Day 1 prior to infusion of IV abatacept, at 30 and 60 minutes after IV infusion of abatacept on Day 1, and at all office visits prior to SC injection of abatacept. Heart rate was also assessed 7 days after the last injection of abatacept for participants who were withdrawn prematurely.
Time Frame: Days 1, 15, 29, 57, 78, and 85
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | ABA [LI]
Number analyzed (Participants) | 167
bpm
  Day 1 HR before infusion (n=167) | 73.9 (9.78)
  Day 15 HR before injection (n=160) | 76.0 (7.91)
  Day 29 HR before injection (n=166) | 75.5 (9.03)
  Day 57 HR before injection (n=164) | 75.5 (8.95)
  Day 78 HR before injection (n=158) | 75.1 (7.78)
  Day 85 HR before injection (n=160) | 74.7 (8.64)

31. Secondary Outcome: LI Period; Mean Temperature (T)
Description: Temperature was taken in participants while seated and measured in degrees celsius. Temperature was assessed at screening, at baseline on Day 1 prior to infusion of IV abatacept, at 30 and 60 minutes after IV infusion of abatacept on Day 1, and at all office visits prior to SC injection of abatacept. Temperature was also assessed 7 days after the last injection of abatacept for participants who were withdrawn prematurely.
Time Frame: Days 1, 15, 29, 57, 78, and 85
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | ABA [LI]
Number analyzed (Participants) | 167
degrees Celsius
  Day 1 T before infusion (n=167) | 36.39 (0.387)
  Day 15 T before injection (n=160) | 36.34 (0.351)
  Day 29 T before injection (n=166) | 36.39 (0.371)
  Day 57 T before injection (n=164) | 36.38 (0.329)
  Day 78 T before injection (n=158) | 36.33 (0.333)
  Day 85 T before injection (n=160) | 36.35 (0.368)

32. Secondary Outcome: DBW; Number of Participants With Death, Serious SAEs, Related SAEs, SAEs Leading to Discontinuation, AEs, Related AEs, or AEs Leading to Discontinuation
Description: as for outcome 23
Time Frame: From Day 85 through Day 169, up to 56 days post last dose in DBW Period or up to first dose in RI Period, whichever occurred earlier
Population: Participants who received at least 1 dose of study medication in DBW period
Measure: Number; unit: participants
Arm/Group | ABA [DBW] | Placebo (PLA) [DBW]
Number analyzed (Participants) | 40 | 80
participants
  Deaths | 0 | 2
  SAEs | 0 | 2
  Related SAEs | 0 | 0
  AEs Leading to Discontinuation | 0 | 0
  AEs | 13 | 29
  Related AEs | 2 | 9
  AEs Leading to Discontinuation | 0 | 0

33. Secondary Outcome: DBW; Number of Participants With AEs of Special Interest
Description: as for outcome 24
Time Frame: as for outcome 32
Population: Participants who received at least 1 dose of study medication in DBW period
Measure: Number; unit: participants
Arm/Group | ABA [DBW] | Placebo (PLA) [DBW]
Number analyzed (Participants) | 40 | 80
participants
  Infections and infestations | 5 | 7
  Malignancies | 0 | 0
  Autoimmune disorders (prespecified) | 0 | 0
  Acute infusional events (prespecified) | 0 | 0
  Peri-infusional events (prespecified) | 0 | 0
  Local injection site reactions (prespecified) | 0 | 0
  Systemic injection reactions (prespecified) | 1 | 1

34. Secondary Outcome: DBW; Number of Participants With Hematology Values Meeting the Marked Abnormality Criteria
Description: Marked abnormality criteria are: Hemoglobin (HGB): >3 g/dL decrease from BL; Hematocrit: <0.75 * BL; Erythrocytes: <0.75 * BL; Platelets (PLT): <0.67 * LLN/>1.5 * ULN, or if BL < LLN then use <0.5 * BL and <100,000 mm^3; Leukocytes: <0.75 * LLN/ >1.25 * ULN, or if BL<LLN then use <0.8 * BL or >ULN, or if BL>ULN then use >1.2 * BL or <LLN; neutrophils+bands: <1.0 * 10^3 cells/uL; eosinophils: >0.750 * 10^3 cells/uL; basophils: > 400 mm^3; monocytes: >2000 mm^3; lymphocytes: <0.750 * 10^3 cells/uL/ >7.50 * 10^3 cells/uL.
Time Frame: as for outcome 32
Population: Participants who received at least 1 dose of study medication in DBW period. N=Number of Participants Analyzed. n (when indicated)= number of participants with data available during the DBW period.
Measure: Number; unit: participants
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 80
participants
  Low HGB (n=40, n=80) | 0 | 0
  Low hematocrit (n=39, n=79) | 0 | 0
  Low erythrocytes (n=40, n=80) | 0 | 0
  Low PLT (n=40, n=80) | 0 | 0
  High PLT (n=40, n=80) | 0 | 0
  Low leukocytes (n=40, n=80) | 0 | 1
  High leukocytes (n=40, n=80) | 0 | 0
  Low neutrophils+bands (n=40, n=80) | 0 | 0
  High eosinophils (n=40, n=80) | 0 | 2
  High basophils (n=40, n=80) | 0 | 0
  High monocytes (n=40, n=80) | 0 | 0
  Low lymphocytes (n=40, n=80) | 2 | 4
  High lymphocytes (n=40, n=80) | 0 | 0

35. Secondary Outcome: DBW; Number of Participants With Liver and Kidney Function Values Meeting the Marked Abnormality Criteria
Description: as for outcome 26
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 80
participants
  High ALP | 0 | 0
  High AST | 0 | 0
  High ALT | 1 | 0
  High GGT | 2 | 0
  High bilirubin | 0 | 0
  High BUN | 0 | 0
  High creatinine | 0 | 1

36. Secondary Outcome: DBW; Number of Participants With Electrolytes Values Meeting the Marked Abnormality Criteria
Description: as for outcome 27
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 80
participants
  Low Na | 0 | 0
  High Na | 0 | 0
  Low K | 0 | 0
  High K | 0 | 0
  Low Cl | 0 | 0
  High Cl | 0 | 0
  Low Ca | 0 | 0
  High Ca | 0 | 0
  Low P | 0 | 0
  High P | 0 | 0

37. Secondary Outcome: DBW; Number of Participants With Other Chemistry and Urinalysis Values Meeting the Marked Abnormality Criteria
Description: MA criteria: serum glucose (Glu): <65 mg/dL/>220 mg/dL;fasting serum Glu: <0.8* LLN/>1.5*ULN,or if BL<LLN then use 0.8*BL or >ULN,or if BL>ULN then use >2.0*BL or <LLN;total protein: <0.9*LLN/>1.1*ULN,or if BL<LLN then use <0.9*BL or >UNL,or if BL>UNL then use >1.1*BL or <LLN; albumin: <0.9*LLN,or if BL<LLN then use <0.75 BL;uric acid: >1.5*ULN,or if BL>ULN then use >2*BL. Urinalysis (Urine protein,urine Glu,urine blood,leukocyte esterase,Red Blood Cells [RBCs], White Blood Cells [WBCs]):Use ≥2 when BL value missing or when pre-dose=0 or 0.5; use ≥3 when pre-dose=1, use ≥4 when pre-dose=2 or 3
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 80
participants
  Low Glu (n=40, n=80) | 2 | 5
  High Glu (n=40, n=80) | 1 | 3
  Low fasting Glu (n=27, n=51) | 0 | 1
  High fasting Glu (n=27, n=51) | 0 | 1
  Low total protein (n=40, n=80) | 0 | 0
  High total protein (n=40, n=80) | 0 | 0
  Low albumin (n=40, n=80) | 0 | 0
  High uric acid (n=40, n=80) | 0 | 0
  High urine protein (n=40, n=80) | 1 | 0
  High urine Glu (n=40, n=80) | 0 | 1
  High urine blood (n=40, n=80) | 3 | 10
  High leukocyte esterase (n=10, n=21) | 1 | 4
  High urine RBC (n=13, n=23) | 1 | 5
  High urine WBC (n=15, n=28) | 6 | 12

38. Secondary Outcome: DBW; Mean Seated Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) During Double Blind Period
Description: Blood pressures were taken in participants while seated, just prior to study drug injection, and measured in millimeters of mercury (mmHg).
Time Frame: Days 113, 141, and 169
Population: Participants who received at least 1 dose of study medication in DBW period. N=Number of Participants Analyzed. n (when indicated)= number of participants with data available at that time point.
Measure: Mean (Standard Deviation); unit: mm mercury (Hg)
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 80
mm mercury (Hg)
  Day 113 SBP before injection (n=39, n=78) | 119.4 (13.29) | 120.4 (15.60)
  Day 141 SBP before injection (n=39, n=76) | 120.3 (12.73) | 121.2 (14.98)
  Day 169 SBP before injection (n=40, n=80) | 119.6 (13.87) | 119.4 (14.11)
  Day 113 DBP before injection (n=39, 78) | 74.2 (10.44) | 74.4 (9.34)
  Day 141 DBP before injection (n=39, n=76) | 76.3 (10.46) | 76.0 (10.60)
  Day 169 DBP before injection (n=40, n=80) | 74.0 (9.51) | 74.7 (8.94)

39. Secondary Outcome: DBW Period; Mean Heart Rate (HR) During Period 2
Description: Heart Rate was taken in participants while seated, just prior to study drug injection, and measured in beats per minute (bpm)
Time Frame: Days 113, 141, and 169
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 80
beats per minute (bpm)
  Day 113 HR before injection (n=40, n=78) | 75.8 (8.07) | 73.9 (8.39)
  Day 141 HR before injection (n=39, n=76) | 75.9 (9.35) | 74.5 (8.45)
  Day 169 HR before injection (n=40, n=80) | 73.8 (8.19) | 74.2 (8.50)

40. Secondary Outcome: DBW Period; Mean Temperature (T) During Period II
Description: Participants were seated and temperature taken just prior to study drug injection.
Time Frame: Days 113, 141, and 169
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | ABA [DBW] | PLA [DBW]
Number analyzed (Participants) | 40 | 80
degrees Celsius
  Day 113 T before infusion (n=40, n=78) | 36.34 (0.488) | 36.44 (0.370)
  Day 141 T before injection (n=39, n=76) | 36.31 (0.355) | 36.36 (0.347)
  Day 169 T before injection (n=40, n=80) | 36.38 (0.364) | 36.32 (0.373)

41. Secondary Outcome: RI; Number of Participants With Death, Serious Adverse Events (SAEs), Related SAEs, SAEs Leading to Discontinuation, AEs, Related AEs, or AEs Leading to Discontinuation
Description: as for outcome 23
Time Frame: From Day 169 through Day 253, up to 56 days post last dose in RI Period or up to first dose in LTE, whichever occurred earlier.
Population: Participants who received at least 1 dose of study medication in RI period.
Measure: Number; unit: participants
Arm/Group | ABA With IV PLA Loading Dose [RI] | PLA Switched to ABA With ABA IV Loading Dose [RI] | PLA Switched to ABA With PLA IV Loading Dose [RI]
Number analyzed (Participants) | 40 | 35 | 44
participants
  Deaths | 0 | 0 | 0
  SAEs | 0 | 0 | 1
  Related SAEs | 0 | 0 | 0
  SAEs Leading to Discontinuation | 0 | 0 | 0
  AEs | 15 | 17 | 16
  Related AEs | 1 | 4 | 4
  AEs Leading to Discontinuation | 0 | 0 | 0

42. Secondary Outcome: RI; Number of Participants With AEs of Special Interest
Description: as for outcome 24
Time Frame: as for outcome 41
Population: Participants who received at least 1 dose of study medication in RI period.
Measure: Number; unit: participants
Arm/Group | ABA With IV PLA Loading Dose [RI] | PLA Switched to ABA With ABA IV Loading Dose [RI] | PLA Switched to ABA With PLA IV Loading Dose [RI]
Number analyzed (Participants) | 40 | 35 | 44
participants
  Infections and infestations | 7 | 8 | 7
  Malignancies | 0 | 0 | 0
  Autoimmune disorders (prespecified) | 0 | 0 | 0
  Acute infusional events (prespecified) | 0 | 0 | 0
  Peri-infusional events (prespecified) | 0 | 0 | 1
  Local injection site reactions (prespecified) | 0 | 0 | 0
  Systemic injection reactions (prespecified) | 0 | 0 | 1

43. Secondary Outcome: RI; Number of Participants With Hematology Values Meeting the Marked Abnormality Criteria
Description: as for outcome 34
Time Frame: as for outcome 41
Population: Participants who received at least 1 dose of study medication in RI period. N=Number of Participants Analyzed. n (when indicated)= number of participants with data available during the RI period.
Measure: Number; unit: participants
Arm/Group | ABA With IV PLA Loading Dose [RI] | PLA Switched to ABA With ABA IV Loading Dose [RI] | PLA Switched to ABA With PLA IV Loading Dose [RI]
Number analyzed (Participants) | 40 | 35 | 44
participants
  Low HGB | 0 | 0 | 0
  Low hematocrit | 0 | 0 | 0
  Low erythrocytes | 0 | 0 | 0
  Low PLT | 0 | 0 | 0
  High PLT | 0 | 0 | 0
  Low leukocytes | 0 | 0 | 0
  High leukocytes | 0 | 1 | 0
  Low neutrophils+bands | 0 | 0 | 0
  High eosinophils | 0 | 0 | 0
  High basophils | 0 | 0 | 0
  High monocytes | 0 | 0 | 0
  Low lymphocytes | 2 | 0 | 0
  High lymphocytes | 0 | 0 | 0

44. Secondary Outcome: RI; Number of Participants With Liver and Kidney Function Values Meeting the Marked Abnormality Criteria
Description: as for outcome 26
Time Frame: as for outcome 41
Population: as for outcome 43
Measure: Number; unit: participants
Arm/Group | ABA With IV PLA Loading Dose [RI] | PLA Switched to ABA With ABA IV Loading Dose [RI] | PLA Switched to ABA With PLA IV Loading Dose [RI]
Number analyzed (Participants) | 40 | 35 | 44
participants
  High ALP | 0 | 0 | 0
  High AST | 0 | 0 | 0
  High ALT | 2 | 0 | 0
  High GGT | 1 | 0 | 0
  High bilirubin | 0 | 0 | 0
  High BUN | 0 | 0 | 0
  High creatinine | 0 | 0 | 0

45. Secondary Outcome: RI; Number of Participants With Electrolytes Values Meeting the Marked Abnormality Criteria
Description: as for outcome 27
Time Frame: as for outcome 41
Population: as for outcome 43
Measure: Number; unit: participants
Arm/Group | ABA With IV PLA Loading Dose [RI] | PLA Switched to ABA With ABA IV Loading Dose [RI] | PLA Switched to ABA With PLA IV Loading Dose [RI]
Number analyzed (Participants) | 40 | 35 | 44
participants
  Low Na | 0 | 0 | 0
  High Na | 0 | 0 | 0
  Low K | 0 | 0 | 1
  High K | 0 | 0 | 0
  Low Cl | 0 | 0 | 0
  High Cl | 0 | 0 | 0
  Low Ca | 0 | 0 | 0
  High Ca | 0 | 0 | 0
  Low P | 0 | 1 | 0
  High P | 0 | 0 | 0

46. Secondary Outcome: RI; Number of Participants With Other Chemistry and Urinalysis Values Meeting the Marked Abnormality Criteria
Description: as for outcome 37
Time Frame: as for outcome 41
Population: as for outcome 43
Measure: Number; unit: participants
Arm/Group | ABA With IV PLA Loading Dose [RI] | PLA Switched to ABA With ABA IV Loading Dose [RI] | PLA Switched to ABA With PLA IV Loading Dose [RI]
Number analyzed (Participants) | 40 | 35 | 44
participants
  Low Glu (n=40, n=35, n=44) | 1 | 1 | 1
  High Glu (n=40, n=35, n=44) | 0 | 1 | 0
  Low fasting Glu (n=27, n=20, n=28) | 1 | 0 | 0
  High fasting glucose (n=27, n=20, n=28) | 0 | 0 | 0
  Low total protein (n=40, n=35, n=44) | 0 | 0 | 0
  High total protein (n=40, n=35, n=44) | 0 | 0 | 0
  Low albumin (n=40, n=35, n=44) | 0 | 0 | 0
  High uric acid (n=40, n=35, n=44) | 0 | 0 | 0
  High urine protein (n=40, n=35, n=44) | 0 | 0 | 1
  High urine glucose (n=40, n=34, n=44) | 0 | 0 | 0
  High urine blood (n=40, n=35, n=44) | 6 | 4 | 7
  High leukocyte esterase (n=14, n=8, n=7) | 4 | 2 | 1
  High urine RBC (n=17, n=14, n=15) | 6 | 3 | 6
  High urine WBC (n=19, n=15, n=15) | 6 | 5 | 4

47. Secondary Outcome: RI Period; Mean Seated Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) During Period III
Time Frame: Days 169, 197, 225, and 253
Population: Participants who received at least 1 dose of study medication in RI period. N=Number of Participants Analyzed. n (when indicated)= number of participants with data available at that time point.
Measure: Mean (Standard Deviation); unit: mm mercury (Hg)
Arm/Group | ABA With IV PLA Loading Dose [RI] | PLA Switched to ABA With ABA IV Loading Dose [RI] | PLA Switched to ABA With PLA IV Loading Dose [RI]
Number analyzed (Participants) | 40 | 35 | 44
mm mercury (Hg)
  Day 169 SBP before infusion (n=39, n=35, n=44) | 121.3 (15.81) | 116.6 (14.78) | 118.9 (13.32)
  Day 197 SBP before injection (n=40, n=35, n=43) | 119.1 (14.07) | 118.4 (15.62) | 121.0 (14.45)
  Day 225 SBP before injection (n=40, n=35, n=42) | 117.8 (14.19) | 118.8 (16.55) | 121.0 (16.88)
  Day 253 SBP before injection (n=40, 35, n=43) | 118.3 (15.00) | 116.1 (14.86) | 120.3 (16.01)
  Day 169 DBP before infusion (n=39, n=35, n=44) | 74.7 (10.46) | 73.5 (9.61) | 74.9 (9.15)
  Day 197 DBP before injection (n=40, n=35, n=43) | 72.9 (9.24) | 71.6 (7.66) | 74.9 (9.51)
  Day 225 DBP before injection (n=40, n=35, n=42) | 73.6 (10.56) | 73.7 (7.84) | 75.5 (10.65)
  Day 253 DBP before injection (n=40, n=35, n=44) | 74.7 (11.24) | 71.5 (9.92) | 76.3 (11.02)

48. Secondary Outcome: RI Period; Mean Heart Rate (HR) During Period III
Time Frame: Days 169, 197, 225, and 253
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | ABA With IV PLA Loading Dose [RI] | PLA Switched to ABA With ABA IV Loading Dose [RI] | PLA Switched to ABA With PLA IV Loading Dose [RI]
Number analyzed (Participants) | 40 | 35 | 44
beats per minute (bpm)
  Day 169 HR before infusion (n=40, n=35, n=44) | 73.4 (8.54) | 73.8 (10.13) | 74.1 (9.35)
  Day 197 HR before injection (n=40, n=35, n=43) | 73.1 (7.52) | 75.1 (7.25) | 70.9 (8.87)
  Day 225 HR before injection (n=40, n=35, n=42) | 73.2 (7.0) | 73.9 (7.43) | 73.2 (7.60)
  Day 253 HR before injection (n=40, n=35, n=43) | 73.6 (8.53) | 74.4 (7.87) | 74.3 (9.36)

49. Secondary Outcome: RI Period; Mean Temperature (T) During Period III
Time Frame: Days 169, 197, 225, and 253
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | ABA With IV PLA Loading Dose [RI] | PLA Switched to ABA With ABA IV Loading Dose [RI] | PLA Switched to ABA With PLA IV Loading Dose [RI]
Number analyzed (Participants) | 40 | 35 | 44
degrees Celsius
  Day 169 T before infusion (n=40, n=35, n=44) | 36.32 (0.423) | 36.29 (0.473) | 36.26 (0.396)
  Day 197 T before injection (n=40, n=35, n=43) | 36.39 (0.405) | 36.37 (0.424) | 36.35 (0.354)
  Day 225 T before injection (n=40, n=35, n=42) | 36.27 (0.375) | 36.38 (0.444) | 36.36 (0.320)
  Day 253 T before injection (n=40, n=34, n=42) | 36.28 (0.473) | 36.32 (0.587) | 36.33 (0.383)

50. Secondary Outcome: Short Term; Abatacept Serum Concentration by Immunogenicity Status as Measured by ELISA by RI Treatment Groups
Description: Pharmacokinetics is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. Cmin=minimum observed plasma concentration of single-dose abatacept. Cmin for each participant was listed by study visit and immunogenicity status (seropositive vs. seronegative) was determined by ELISA.
Time Frame: Day 197 through Day 253
Population: Participants treated during the RI Period with at least 1 immunogenicity result (ELISA) during this period. N=Number of Participants Analyzed, n=number of participants with data for that time point
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | ABA With IV PLA Loading Dose [RI] | PLA Switched to ABA With ABA IV Loading Dose [RI] | PLA Switched to ABA With PLA IV Loading Dose [RI]
Number analyzed (Participants) | 40 | 35 | 44
ug/mL
  Day 197 seropositive (n=2, n=1, n=1) | 39.17 (10.510) | 33.73 (NA) — Standard deviation not applicable for 1 participant. | 18.05 (NA) — Standard deviation not applicable for 1 participant.
  Day 197 seronegative (n=33, n=32, n=40) | 34.45 (10.578) | 35.67 (10.365) | 22.76 (8.740)
  Day 225 seropositive (n=0, n=1, n=1) | NA (NA) — Data not measured/analyzed for 0 participants. | 34.18 (NA) — Standard deviation not applicable for 1 participant. | 21.69 (NA) — Standard deviation not applicable for 1 participant.
  Day 225 seronegative (n=36, n=29, n=41) | 27.86 (9.514) | 31.70 (10.635) | 29.24 (13.897)
  Day 253 seropositive (n=1, n=0, n=2) | 29.49 (NA) — Standard deviation no applicable for 1 participant. | NA (NA) — Data not measured/analyzed for 0 participants. | 26.23 (0.776)
  Day 253 seronegative (n=34, n=30, n=39) | 30.17 (9.856) | 28.26 (10.211) | 26.80 (10.547)

51. Secondary Outcome: Short Term; Abatacept Serum Concentration by Immunogenicity Status as Measured by ECL by RI Treatment Groups
Description: Pharmacokinetics is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. Cmin=minimum observed plasma concentration of single-dose abatacept. Cmin for each participant was listed by study visit and immunogenicity status (seropositive vs. seronegative) was determined by ECL.
Time Frame: Day 197 through Day 253
Population: Participants treated in RI period with at least 1 immunogenicity result (ECL) during RI period. N=Number of Participants Analyzed, n=number of participants with data for that time point
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | ABA With IV PLA Loading Dose [RI] | PLA Switched to ABA With ABA IV Loading Dose [RI] | PLA Switched to ABA With PLA IV Loading Dose [RI]
Number analyzed (Participants) | 40 | 35 | 44
ug/mL
  Day 197 seropositive (n=0, n=0, n=0) | NA (NA) — Data not measured/analyzed for 0 participants. | NA (NA) — Data not measured/analyzed for 0 participants. | NA (NA) — Data not measured/analyzed for 0 participants.
  Day 197 seronegative (n=35, n=33, n=41) | 34.72 (10.479) | 35.61 (10.207) | 22.65 (8.662)
  Day 225 seropositive (n=0, n=0, n=0) | NA (NA) — Data not measured/analyzed for 0 participants. | NA (NA) — Data not measured/analyzed for 0 participants. | NA (NA) — Data not measured/analyzed for 0 participants.
  Day 225 seronegative (n=36, n=30, n=42) | 27.86 (9.514) | 31.79 (10.460) | 29.06 (13.776)
  Day 253 seropositive (n=0, n=0, n=0) | NA (NA) — Data not measured/analyzed for 0 participants. | NA (NA) — Data not measured/analyzed for 0 participants. | NA (NA) — Data not measured/analyzed for 0 participants.
  Day 253 seronegative (n=36, n=30, n=42) | 29.75 (9.872) | 28.26 (10.211) | 26.28 (10.645)

52. Secondary Outcome: ST; Number of Participants Positive for Anti-nuclear Antibody (ANA), Anti-double Stranded DNA Antibody (dsDNA), or Rheumatoid Factor (RF) at Day 253 According to Baseline Status (Negative at Baseline or Positive at Baseline) by DBW Treatment Groups
Description: Venous blood was collected and tested for anti-nuclear antibodies, anti-dsDNA antibodies, and rheumatoid factor. ANA were detected by means of immunofluorescent antibodies. An anti-DNA radioimmunoassay was used for detection of anti-dsDNA antibodies (Diagnostic Products Corporation). RF was measured by an immunoturbidimetric assay (Roche Tina-Quant). Determinations of antibody or RF status were made at baseline and Day 253.
Time Frame: Baseline, Day 253
Population: Participants treated in DBW period with at least 1 immunogenicity result (immunofluorescence, radioimmunoassay, or immunoturbidimetry) during this period. N=Number of Participants Analyzed, n=number of participants with data for that time point
Measure: Number; unit: participants
Arm/Group | ABA [DBW] | Placebo (PLA) [DBW]
Number analyzed (Participants) | 40 | 79
participants
  BL ANA negative (n=27, n=57) | 1 | 3
  BL ANA positive (n=11, 18) | 5 | 10
  BL dsDNA negative (n=33, n=63) | 1 | 2
  BL dsDNA positive (n=3, n=6) | 2 | 3
  BL RF negative (n=6, n=10) | 0 | 0
  BL RF positive (n=34, n=64) | 34 | 63

53. Secondary Outcome: LTE: DAS28-CRP Mean Change From Baseline (Day 1) Over Time - All Participants Treated in LTE
Description: DAS28=continuous disease measure composite of 4 variables: number of tender joints out of 28, number of swollen joints out of 28, level of serum reactant protein CRP, and participant global assessment of disease activity measured on a visual analogue scale. DAS28-CRP has numeric thresholds defining high disease activity (> 5.1), low disease activity (≤ 3.2) and remission (< 2.6). Last day of ST is Day 85 for Period I Nonresponders and Day 253 for ST Completers . Data are not available(NA) for the period from Day 113 to Day 253 for Period 1 non-responders. Note: Day 85 and Day 337 assessments for the Period I Nonresponder cohort in fact represent consecutive assessments with an interval of approximately 1 month. For Period I nonresponder, study days do not represent treatment days. Study Day 337 for a Period I nonresponder actually corresponds to that participant's Treatment Day 169.
Time Frame: For Period 1 non-responders: as of Study Day 85 and up to Day 1821. For ST completers: as of Study Day 253 and up to Day 1821.
Population: The LTE Treated Population contained those participants who received at least 1 dose of study medication during the LTE. Participants in LTE either completed Period 3 or were nonresponders at the end of Period 1. n=number of participants with both baseline and post-baseline measurements.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- LTE Abatacept for LI Period 1 Non-responders: Participants received Abatacept SC injections (fixed dose of 125 mg) during Lead-in (LI) Period 1 for 12 weeks. If after 12 weeks the participant was a non-responder (unable to achieve DAS28-CRP decrease by ≥ 0.6 from Day 1), they directly entered the LTE receiving open label Abatacept SC injections (125 mg) starting on Day 85 and weekly for 12 weeks (ie, participants did not enter DBW or RI periods). If clinical response was achieved, participant continued in LTE until SC administration of Abatacept was approved by the respective country and commercially available or until sponsor elected to terminate the study.
- LTE Abatacept for Short Term Completers: Participant's who successfully completed the Short Term of the study, entered the LTE on Day 253 and received weekly open-label SC abatacept (125 mg) in the LTE until SC administration of ABA was approved by the respective country and commercially available or until the sponsor elected to terminate the study. Participants who completed the ST study (Completers) had received ABA during LI Period 1, entered DBW Period 2 (ABA or PLA), and in RI Period 3 continued/switched to ABA (with either ABA or PLA IV loading dose, as appropriate).
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 36 | 113
units on a scale
  Study Day 15; Treatment Day 15 (n=31, 106) | -0.48 (0.14) | -0.79 (0.06)
  Study Day 85; Treatment Day 85 (n=36, 112) | -0.35 (0.21) | -1.91 (0.09)
  Study Day 253; Treatment Day 85 (n=0, n=109) | NA (NA) — No data collected. 0 participants available. Period 1 non-responders started LTE on Study Day 85, not Study Day 253. | -2.29 (0.09)
  Study Day 337; Treatment Day 169 (n=34,n=113) | -1.51 (0.16) | -2.34 (0.09)
  Study Day 365; Treatment Day 197 (n=31, n=110) | -1.83 (0.19) | -2.23 (0.10)
  Study Day 533; Treatment Day 365 (n=32, n=106) | -1.86 (0.19) | -2.28 (0.12)
  Study Day 729; Treatment Day 561 (n=30, n=106 | -1.81 (0.19) | -2.16 (0.12)
  Study Day 1093; Treatment Day 925 (n=26, n=98) | -1.94 (0.18) | -2.12 (0.12)
  Study Day 1261; Treatment Day 1093 (n=25, n=96) | -1.70 (0.15) | -2.20 (0.13)
  Study Day 1821; Treatment Day 1653 (n=20, n=67) | -1.86 (0.20) | -2.55 (0.14)

54. Secondary Outcome: LTE: Percent of Participants Who Achieved Clinical Remission in the Long Term Extension - All Participants Treated in LTE
Description: DAS28=continuous disease measure composite of 4 variables: number of tender joints out of 28, number of swollen joints out of 28, level of serum reactant protein CRP, and participant global assessment of disease activity measured on a visual analogue scale. Clinical remission=DAS28-CRP score<2.6. Percent=Number of participants meeting remission divided by number of participants evaluated. Last day of ST is Day 85 for Period I Nonresponders and Day 253 for ST Completers . Data are not available (NA) for the period from Day 113 to Day 253 for Period 1 non-responders. Note: Day 85 and Day 337 assessments for the Period I Nonresponder cohort in fact represent consecutive assessments with an interval of approximately 1 month. For Period I nonresponder, study days do not represent treatment days. Study Day 337 for a Period I nonresponder actually corresponds to that participant's Treatment Day 169.
Time Frame: For Period I non-responders: as of Study Day 85 and up to Study Day 1821. For ST completers: as of Study Day 253 and up to Study Day 1821
Population: The LTE Treated Population contained those participants who received at least 1 dose of study medication during the LTE. Participants in LTE either completed Period 3 or were nonresponders at the end of Period 1. n= number of participants evaluated at each specific timepoint
Measure: Number; unit: percentage of participants
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 36 | 113
percentage of participants
  Study Day 85 (n=36, n=112) | 11.1 | 36.6
  Study Day 253 (n=0, n=109) | NA — no data available. 0 participants. Period 1 non-responders entered LTE on Study Day 85, not Study Day 253. | 59.6
  Study Day 337 (n=34, n=113) | 50.0 | 59.3
  Study Day 729 (n=30, n=106) | 53.3 | 54.7
  Study Day 1093 (n=26, 90) | 73.1 | 51.0
  Study Day 1261 (n=25, n=96) | 48.0 | 59.4
  Study Day 1821 (n=20, n=67) | 60.0 | 59.7

55. Secondary Outcome: LTE: Percent of Participants With Low Disease Activity in Long Term Extension: All Participants Treated in LTE
Description: DAS28:continuous disease measure composite of 4 variables: number of tender joints out of 28 joints, number of swollen joints out of 28 joints, level of the serum reactant protein CRP, and participant global assessment of disease activity measure on a visual analogue scale. Low disease activity score: ≤ 3.2. Percent=Number of participants with Low Disease Activity divided by number of participants evaluated. Last day of ST is Day 85 for Period I Nonresponders and Day 253 for ST Completers . Data are not available(NA) for the period from Day 113 to Day 253 for Period 1 non-responders. Note: Day 85 and Day 337 assessments for the Period I Nonresponder cohort in fact represent consecutive assessments with an interval of approximately 1 month. For Period I nonresponder, study days do not represent treatment days. Study Day 337 for a Period I nonresponder actually corresponds to that participant's Treatment Day 169.
Time Frame: as for outcome 53
Population: The LTE Treated Population contained those participants who received at least 1 dose of study medication during the LTE. Participants in LTE either completed Period 3 or were nonresponders at the end of Period 1.
Measure: Number; unit: percentage of participants
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 36 | 113
percentage of participants
  Study Day 85 (n=36, n=112) | 27.8 | 66.1
  Study Day 253 (n=0, n=109) | NA — no data available. 0 participants. Period 1 non-responders entered LTE on Study Day 85, not Study Day 253. | 75.2
  Study Day 337 (n=34, n=113) | 67.6 | 76.1
  Study Day 729 (n=30, n=106) | 73.3 | 73.6
  Study Day 1093 (n=26, n=98) | 80.8 | 67.3
  Study Day 1261 (n=25, n=96) | 68.0 | 75.0
  Study Day 1821 (n=20, n=67) | 80.0 | 88.1

56. Secondary Outcome: LTE: Percent of Participants With HAQ Response Over Time - All Participants Treated in LTE
Description: The disability section of the full HAQ includes 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. The questions are evaluated on a 4-point scale: 0=without any difficulty, 1= with some difficulty, 2= with much difficulty, and 3= unable to do. Higher scores= greater dysfunction. A disability index (DI) was calculated by summing the worst scores in each domain and dividing by the number of domains answered. Clinically meaningful HAQ response=an improvement of at least 0.3 units from baseline in HAQ DI. Percent=number of participants with HAQ response divided by number of participants in the analysis. Since Period I Non-responders proceeded directly to the LTE at the end of Period I (Day 85), study days do not represent treatment days.
Time Frame: Study Days 1 (Baseline),15, 29, 57, 78, 85, 253, 337, 365, 449, 533, 617, 729, 813, 897, 981, 1093, 1177, 1261, 1345, 1457, 1541,1625,1709,1821,1905,1989, 2073
Population: The LTE Treated Population contained those participants who received at least 1 dose of study medication during the LTE. Participants in LTE either completed Period 3 or were non-responders at the end of Period 1. n= number of participants with data who were evaluated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 37 | 113
percentage of participants
  Study Day 15; Treatment Day 15 (n=34, n=110) | 20.6 [7.0 to 34.2] | 44.5 [35.3 to 53.8]
  Study Day 29; Treatment Day 29 (n=36, n=113) | 27.8 [13.1 to 42.4] | 56.6 [47.5 to 65.8]
  Study Day 57; Treatment Day 57 (n=36, n=112) | 44.4 [28.2 to 60.7] | 64.3 [55.4 to 73.2]
  Study Day 78; Treatment Day 78 (n=34, n=103) | 41.2 [24.6 to 57.7] | 68.0 [58.9 to 77.0]
  Study Day 85; Treatment Day 85 (n=37, n=112) | 40.5 [24.7 to 56.4] | 74.1 [66.0 to 82.2]
  Study Day 253; Treatment Day 85 (n=0, n=109) | NA [NA to NA] — no data collected. 0 participants. Period 1 non-responders entered LTE on Study Day 85 not Study Day 253. | 78.0 [70.2 to 85.8]
  Study Day 337; Treatment Day 169 (n=34, n=113) | 50.0 [33.2 to 66.8] | 79.6 [72.2 to 87.1]
  Study Day 365; Treatment Day 197 (n=32, n=111) | 53.1 [35.8 to 70.4] | 78.4 [70.7 to 86.0]
  Study Day 449; Treatment Day 281 (n=32, n=109) | 56.3 [39.1 to 73.4] | 73.4 [65.1 to 81.7]
  Study Day 533; Treatment Day 365 (n=32, n=108) | 59.4 [42.4 to 76.4] | 72.2 [63.8 to 80.7]
  Study Day 617; Treatment Day 449 (n=31, n=107) | 54.8 [37.3 to 72.4] | 70.1 [61.4 to 78.8]
  Study Day 729; Treatment Day 561 (n=30, n=107) | 60.0 [42.5 to 77.5] | 70.1 [61.4 to 78.8]
  Study Day 813; Treatment Day 645 (n=30, n=106) | 53.3 [35.5 to 71.2] | 71.7 [63.1 to 80.3]
  Study Day 897; Treatment Day 729 (n=30, n=103) | 50.0 [32.1 to 67.9] | 76.7 [68.5 to 84.9]
  Study Day 981; Treatment Day 813 (n=29, n=100) | 44.8 [26.7 to 62.9] | 73.0 [64.3 to 81.7]
  Study Day 1093; Treatment Day 925 (n=28, n=99) | 50.0 [31.5 to 68.5] | 73.7 [65.1 to 82.4]
  Study Day 1177; Treatment Day 1009 (n=26, n=99) | 61.5 [42.8 to 80.2] | 68.7 [59.6 to 77.8]
  Study Day 1261; Treatment Day 1093 (n=25, n=97) | 60.0 [40.8 to 79.2] | 70.1 [61.0 to 79.2]
  Study Day 1345; Treatment Day 1177 (n=25, n=89) | 64.0 [45.2 to 82.8] | 70.8 [61.3 to 80.2]
  Study Day 1457; Treatment Day 1289 (n=24, n=79) | 66.7 [47.8 to 85.5] | 72.2 [62.3 to 82.0]
  Study Day 1541; Treatment Day 1373 (n=21, n=75) | 61.9 [41.1 to 82.7] | 69.3 [58.9 to 79.8]
  Study Day 1625; Treatment Day 1457 (n=21, n=73) | 52.4 [31.0 to 73.7] | 74.0 [63.9 to 84.0]
  Study Day 1709; Treatment Day 1541 (n=20, n=71) | 60.0 [38.5 to 81.5] | 74.6 [64.5 to 84.8]
  Study Day 1821; Treatment Day 1653 (n=20, n=68) | 65.0 [44.1 to 85.9] | 73.5 [63.0 to 84.0]
  Study Day 1905; Treatment Day 1737 (n=19, n=5) | 63.2 [41.5 to 84.8] | 80.0 [44.9 to 100.0]
  Study Day 1989; Treatment Day 1821 (n=19, n=0) | 68.4 [47.5 to 89.3] | NA [NA to NA] — no data collected due to 0 participant available.
  Study Day 2073; Treatment Day 1905 (n=5, n=0) | 100.0 [100.0 to 100.0] | NA [NA to NA] — no data collected due to 0 participant available.

57. Secondary Outcome: LTE: Overall Percentage of Participants With Positive Anti-Abatacept or Anti-CTLA4 Antibody Responses (ECL Method) for On-Treatment Visits, Post Last Dose Visits, and Overall Study - All Participants Treated in LTE
Description: Serum samples from Abatacept-treated adult participants with active RA were screened for the presence of drug-specific antibodies using electrochemiluminescence (ECL). The percent of participants with a positive abatacept induced immunogenicity response against cytotoxic T-lymphocyte antigen 4 (CTLA4) and possibly immunoglobulin (Ig), or against Ig and/or Junction Region was calculated by number of participants with a positive response divided by number of participants evaluated. Overall for on-treatment includes treatment visits on Days 337, 365, 449, 533, 617, 729, 813, 897, 981, 1093, 1177, 1261, 1457, 1625, 1821, and 1989.
Time Frame: Days 337, 365, 449, 533, 617, 729, 813, 897, 981, 1093, 1177, 1261, 1457, 1625, 1821, 1989 and 28, 56, 85, 168 days post last dose in LTE
Population: All participants treated in LTE period with at least 1 immunogenicity result (ECL) during LTE period. n=number of participants evaluated.
Measure: Number; unit: percentage of participants
Groups:
- LTE Abatacept for All Participants: This group includes all participants who received at least one dose of 125 mg SC Abatacept during the LTE and includes both the LI Period 1 non-responder and the ST Completer cohorts.
Arm/Group | LTE Abatacept for All Participants
Number analyzed (Participants) | 149
percentage of participants
  Overall Study (n=149) | 20.1
  Overall on Treatment Visit Days (n=147) | 15.6
  28 Days post last dose (n=110) | 7.3
  56 Days post last dose (n=16) | 6.3
  85 Days post last dose (n=103) | 7.8
  168 Days post last dose (n=21) | 23.8
  Overall Post Visits (n=126) | 12.7

58. Secondary Outcome: LTE: Number of Participants With Death, Related SAEs, SAEs Leading to Discontinuation, Related AEs, or AEs Leading to Discontinuation During Long Term Extension (LTE)
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event. SAEs include hospitalizations for elective surgical procedures.All deaths reported during the LTE including those that occurred > 56 days after the last dose. Related AE or SAE defined as AE or SAE with Certain, Probable, Possible, or Missing relationship to study medication. All participants who completed the ST period could enter the open label LTE on Day 253; LI Period 1 non-responders could directly enter the LTE.
Time Frame: For Period I non-responders: as of Day 85 and up to completion of LTE (FEB 2014), up to 56 days post last dose. For ST completers: as of Day 253 and up to completion of LTE (FEB 2014) up to 56 days post last dose.
Population: Participants who received at least 1 dose of study medication in LTE period
Measure: Number; unit: participants
Groups:
- LTE Abatacept for Short Term Completers: Participant's who successfully completed the Short Term of the study, could enter the LTE on Day 253 and receive weekly open-label SC abatacept (125 mg) in the LTE until SC administration of ABA was approved by the respective country and commercially available or until the sponsor elected to terminate the study. Participants who completed the ST study (Completers) had received ABA during LI Period 1, entered DBW Period 2 (ABA or PLA), and in RI Period 3 continued/switched to ABA (with either ABA or PLA IV loading dose, as appropriate).
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 37 | 113
participants
  Deaths | 1 | 6
  Related SAEs | 0 | 3
  SAEs Leading to Discontinuation | 1 | 5
  Related AEs | 9 | 45
  AEs Leading to Discontinuation | 2 | 5

59. Secondary Outcome: LTE: Number of Participants With AEs of Special Interest During LTE
Description: AEs of special interest in LTE are those AEs that may be associated with the use of immunomodulatory drugs, including all infections and opportunistic infections; autoimmune disorders; malignancies, local injection site reaction (pre-specified AEs occurring at the site of SC injection) and systemic injection site reactions (pre-specified systemic AEs such as hypersensitivity reactions occurring within 24 hours of SC injection)
Time Frame: For Period I non-responders: as of Day 85 and up to completion of LTE (FEB 2014) up to 56 days post last dose. For ST completers: as of Day 253 and up to completion of LTE (FEB 2014) up to 56 days post last dose.
Population: Participants who received at least 1 dose of study medication in LTE period
Measure: Number; unit: participants
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 37 | 113
participants
  Infections and infestations | 23 | 78
  Malignancies | 1 | 3
  Autoimmune disorders (prespecified) | 3 | 8
  Local injection site reactions (prespecified) | 0 | 3
  Systemic injection reactions (prespecified) | 3 | 11

60. Secondary Outcome: LTE: Number of Participants With Hematology Values Meeting the Marked Abnormality Criteria During LTE
Description: as for outcome 34
Time Frame: For Period I non-responders: as of Day 85 and up to completion of LTE (FEB 2014). For ST completers: as of Day 253 and up to completion of LTE (FEB 2014). Data included up to 56 days post last dose.
Population: Participants who received at least 1 dose of study medication in LTE period and who had data available during the LTE period.
Measure: Number; unit: participants
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 35 | 113
participants
  Low HGB | 1 | 4
  Low hematocrit | 0 | 2
  Low erythrocytes | 0 | 1
  Low PLT | 0 | 1
  Low leukocytes | 1 | 5
  High leukocytes | 0 | 6
  Low neutrophils+bands | 0 | 2
  High eosinophils | 3 | 14
  Low lymphocytes | 5 | 9

61. Secondary Outcome: LTE: Number of Participants With Liver and Kidney Function Values Meeting the Marked Abnormality Criteria During LTE
Description: as for outcome 26
Time Frame: as for outcome 60
Population: as for outcome 60
Measure: Number; unit: participants
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 35 | 113
participants
  High AST | 0 | 3
  High ALT | 2 | 2
  High GGT | 1 | 8
  High bilirubin | 0 | 1
  High BUN | 0 | 7
  High creatinine | 4 | 11

62. Secondary Outcome: LTE: Number of Participants With Electrolyte Values Meeting the Marked Abnormality Criteria During LTE
Description: as for outcome 27
Time Frame: as for outcome 60
Population: as for outcome 60
Measure: Number; unit: participants
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 35 | 113
participants
  High Na | 1 | 0
  Low K | 0 | 3
  High Cl | 1 | 0
  Low P | 0 | 5
  High P | 1 | 0

63. Secondary Outcome: LTE: Number of Participants With Other Chemistry and Urinalysis Values Meeting the Marked Abnormality Criteria During LTE
Description: as for outcome 37
Time Frame: as for outcome 60
Population: Participants who received at least 1 dose of study medication in LTE period. N=Number of Participants Analyzed. n (when indicated)= number of participants with data available during the LTE period.
Measure: Number; unit: participants
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 35 | 113
participants
  Low Glu (n=35, n=113) | 6 | 16
  High Glu (n=35, n=113) | 1 | 6
  Low fasting Glu (n=14, n=75) | 4 | 2
  High fasting Glu (n=14, n=75) | 0 | 6
  Low total protein (n=35, n=113) | 1 | 0
  Low albumin (n=35, n=113) | 1 | 0
  High urine protein (n=35, n=113) | 2 | 11
  High urine Glu (n=35, n=113) | 1 | 3
  High urine blood (n=35, n=113) | 5 | 30
  High urine WBC (n=22, n=81) | 12 | 39
  High urine RBC (n=16, n=66) | 1 | 27
  High leukocyte esterase (n=19, n=67) | 6 | 18

64. Secondary Outcome: LTE: Mean Seated Systolic Blood Pressure (SBP) During LTE
Description: During LTE, blood pressure was taken in participants while seated, measured in millimeters of mercury (mmHg) and were assessed at all office visits prior to SC injection of abatacept. Vital signs were also assessed 7 days after the last injection of abatacept for participants who were withdrawn prematurely.
Time Frame: Days 337, 365, 449, 533, 617, 729,813, 897,981, 1093, 1177,1261,1345, 1457,1541,1625,1709,1821,1905,1989,2073
Population: Participants who received at least 1 dose of study medication in LTE period. N=Number of Participants Analyzed. n (when indicated)= number of participants with data available at that time point.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 35 | 110
mm Hg
  Day 337 (n=35, n=110) | 125.7 (13.76) | 120.8 (15.92)
  Day 365 (n=32, n=108) | 122.7 (14.26) | 120.4 (15.11)
  Day 449 (n=32, n=108) | 122.9 (15.08) | 119.5 (14.88)
  Day 533 (n=32, n=108) | 123.0 (14.48) | 120.7 (15.75)
  Day 617 (n= 30, n=107) | 121.7 (13.26) | 118.7 (15.30)
  Day 729 (n=30, n=106) | 122.2 (11.77) | 121.5 (17.41)
  Day 813 (n=30, n=101) | 126.6 (12.66) | 120.6 (15.65)
  Day 897 (n=30, n=102) | 123.9 (11.92) | 122.5 (14.92)
  Day 981 (n=28, n=100) | 123.3 (12.23) | 122.9 (15.03)
  Day 1093 (n=26, n=99) | 127.2 (18.41) | 123.7 (15.11)
  Day 1177 (n=25, n=96) | 125.8 (11.17) | 123.0 (15.96)
  Day 1261 (n=25, n=92) | 124.9 (11.04) | 119.7 (13.64)
  Day 1345 (n=24, n=82) | 124.5 (13.11) | 121.9 (14.49)
  Day 1457 (n=21, n=79) | 124.1 (14.75) | 125.5 (18.41)
  Day 1541 (n=21, n=79) | 126.1 (15.06) | 122.3 (14.53)
  Day 1625 (n=21, n=77) | 122.4 (9.09) | 120.3 (13.76)
  Day 1709 (n=21, n=74) | 123.0 (13.08) | 121.9 (14.90)
  Day 1821 (n=20, n=33) | 125.4 (13.22) | 124.3 (10.95)
  Day 1905 (n=18, n=0) | 121.8 (13.14) | NA (NA) — No participants; n=0
  Day 1989 (n=13, n=0) | 124.6 (9.56) | NA (NA) — No participants; n=0
  Day 2073 (n=1, n=0) | 113.0 (0) | NA (NA) — No participants; n=0

65. Secondary Outcome: LTE: Mean Seated Diastolic Blood Pressure (DBP) During LTE
Description: as for outcome 64
Time Frame: Days 337, 365, 449, 533, 617, 729,813, 897,981, 1093, 1177,1261, 1345, 1457,1541,1625,1709,1821,1905,1989,2073
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 35 | 110
mmHg
  Day 337 (n=35, 110) | 76.3 (6.69) | 75.4 (11.18)
  Day 365 (n=32, 108) | 75.1 (10.42) | 75.1 (8.94)
  Day 449 (n=32, n=108) | 77.3 (9.48) | 73.8 (9.12)
  Day 533 (n=32, n=108) | 75.5 (8.43) | 75.4 (9.14)
  Day 617 (n=30, n=107) | 74.2 (8.81) | 74.8 (9.45)
  Day 729 (n=30, n=106) | 73.2 (8.42) | 76.1 (9.86)
  Day 813 (n=30, n=101) | 75.7 (9.39) | 76.4 (9.30)
  Day 897 (n=30, n=102) | 76.8 (8.41) | 75.5 (9.09)
  Day 981 (n=28, n=100) | 77.4 (6.55) | 76.1 (9.67)
  Day 1093 (n=26, n=99) | 76.7 (7.11) | 75.9 (9.88)
  Day 1177 (n=25, n=96) | 76.3 (6.32) | 75.9 (8.58)
  Day 1261 (n=25, n=92) | 75.4 (8.18) | 75.6 (8.59)
  Day 1345 (n=24, n=82) | 75.3 (6.08) | 75.6 (9.03)
  Day 1457 (n=21, n=79) | 75.6 (9.18) | 77.1 (10.04)
  Day 1541 (n=21, n=79) | 76.9 (8.14) | 76.0 (9.15)
  Day 1625 (n=21, n=77) | 77.2 (5.89) | 74.9 (9.01)
  Day 1709 (n=21, n=74) | 75.0 (9.47) | 75.4 (9.09)
  Day1821 (n=20, n=33) | 76.0 (7.99) | 78.3 (7.57)
  Day 1905 (n=18, n=0) | 73.2 (7.96) | NA (NA) — No participants; n=0
  Day 1989 (n=13, n=0) | 77.0 (5.31) | NA (NA) — No participants; n=0
  Day 2073 (n=1, n=0) | 69.0 (0) | NA (NA) — No participants; n=0

66. Secondary Outcome: LTE: Mean Heart Rate (HR) During LTE
Description: During LTE, heart rate was taken in participants while seated, measured in beats per minute (bpm) and was assessed at all office visits prior to SC injection of abatacept. Heart rate was also assessed 7 days after the last injection of abatacept for participants who were withdrawn prematurely.
Time Frame: Days 337, 365, 449, 533, 617, 729,813, 897,981, 1093, 1177,1261, 1345, 1457,1541,1625,1709,1821,1905,1989,2073
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 35 | 110
bpm
  Day 337 (n=35, n=110) | 74.3 (7.07) | 74.9 (8.76)
  Day 365 (n=32, n=109) | 74.2 (7.76) | 75.7 (8.45)
  Day 449 (n=32, n=108) | 74.4 (6.62) | 75.7 (7.76)
  Day 533 (n=32, n=108) | 75.8 (6.62) | 74.7 (8.32)
  Day 617 (n=30, n=107) | 75.7 (6.96) | 76.0 (8.35)
  Day 729 (n=30, n=106) | 74.2 (8.60) | 75.1 (8.70)
  Day 813 (n=30, n=103) | 72.4 (7.57) | 76.2 (9.23)
  Day 897 (n=30, n=102) | 76.1 (7.71) | 76.3 (8.15)
  Day 981 (n=28, n=100) | 74.4 (8.00) | 76.5 (10.75)
  Day 1093 (n=26, n=99) | 76.3 (8.35) | 75.0 (9.20)
  Day 1177 (n=25, n=97) | 77.6 (6.89) | 75.3 (9.00)
  Day 1261 (n=25, n=92) | 75.7 (7.97) | 74.4 (8.91)
  Day 1345 (n=24, n=82) | 73.5 (8.54) | 73.6 (8.62)
  Day 1457 (n=21, n=79) | 75.0 (7.67) | 76.8 (7.96)
  Day 1541 (n=21, n=79) | 77.3 (7.34) | 75.1 (8.51)
  Day 1625 (n=21, n=77) | 76.9 (7.77) | 75.2 (8.12)
  Day 1709 (n=21, n=74) | 78.7 (6.86) | 74.7 (8.83)
  Day 1821 (n=20, n=33) | 79.5 (7.80) | 78.2 (6.78)
  Day 1905 (n=18, n=0) | 77.1 (8.97) | NA (NA) — No participants; n=0
  Day 1989 (n= 13, n=0) | 77.2 (9.53) | NA (NA) — No participants; n=0
  Day 2073 (n=1, n=0) | 63.0 (0) | NA (NA) — No participants; n=0

67. Secondary Outcome: LTE: Mean Temperature (T) During LTE
Description: During LTE, temperature was taken in participants while seated, measured in degrees celsius and was assessed at all office visits prior to SC injection of abatacept. Temperature was also assessed 7 days after the last injection of abatacept for participants who were withdrawn prematurely.
Time Frame: Days 337, 365, 449,533, 617, 729,813, 897,981, 1093, 1177,1261, 1345, 1457,1541,1625,1709,1821,1905,1989,2073
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | LTE Abatacept for LI Period 1 Non-responders | LTE Abatacept for Short Term Completers
Number analyzed (Participants) | 35 | 110
degrees Celsius
  Day 337 (n=35, n=110) | 36.29 (0.285) | 36.31 (0.370)
  Day 365 (n=32, n=108) | 36.35 (0.370) | 36.30 (0.393)
  Day 449 (n=32, n=108) | 36.40 (0.354) | 36.30 (0.294)
  Day 533 (n=32, n=108) | 36.42 (0.358) | 36.30 (0.312)
  Day 617 (n=30, n=106) | 36.38 (0.248) | 36.37 (0.316)
  Day 729 (n=30, n=106) | 36.47 (0.252) | 36.27 (0.332)
  Day 813 (n=30, n=103) | 36.49 (0.284) | 36.30 (0.324)
  Day 897 (n=30, n=102) | 36.44 (0.254) | 36.26 (0.325)
  Day 981 (n=28, n=100) | 36.48 (0.259) | 36.30 (0.295)
  Day 1093 (n=26, n=99) | 36.35 (0.370) | 36.28 (0.278)
  Day 1177 (n=25, n=97) | 36.41 (0.277) | 36.24 (0.327)
  Day 1261 (n=25, n=92) | 36.39 (0.256) | 36.24 (0.276)
  Day 1345 (n=24,n=82) | 36.29 (0.285) | 36.23 (0.232)
  Day 1457 (n=21, n=79) | 36.32 (0.253) | 36.23 (0.242)
  Day 1541 (n=21, n=79) | 36.34 (0.223) | 36.24 (0.198)
  Day 1625 (n=21, n=77) | 36.37 (0.215) | 36.20 (0.214)
  Day 1709 (n=21, n=74) | 36.35 (0.178) | 36.24 (0.249)
  Day 1821 (n=20, n=33) | 36.25 (0.315) | 36.26 (0.228)
  Day 1905 (n=18, n=0) | 36.37 (0.211) | NA (NA) — No participants; n=0
  Day 1989 (n=13, n=0) | 36.35 (0.139) | NA (NA) — No participants; n=0
  Day 2073 (n=1, n=0) | 36.40 (0) | NA (NA) — No participants; n=0

ADVERSE EVENTS:
Time Frame: Day 1 up to 56 days post last dose, through LTE (for those participating in LTE); Day 1 up to 56 days post last dose until final day of study for Period 1 non-completers.
Description: Study initiated November 2007 and LTE ended February 2014. Periods 1, 2, 3 were each 12 weeks in length. LTE started Day 253 and continued until abatacept was approved by the respective country and commercially available or until the sponsor elected to terminate the study.
Groups:
- Period 1 Non-Completers: Participants received Abatacept SC injections (fixed dose of 125 mg) during Lead-in (LI) Period 1 for 12 weeks. These participants did not complete the Period and did not continue in the study.
- Period 1 Non-Responders: Participants received Abatacept SC injections (fixed dose of 125 mg) during Lead-in (LI) Period 1 for 12 weeks. If after 12 weeks the participant was a non-responder (unable to achieve DAS28-CRP decrease by ≥ 0.6 from Day 1), they directly entered the LTE receiving open label Abatacept SC injections (125 mg) starting on Day 85 until completion of the LTE.
- Abatacept Received in Period 2: Participants who responded to abatacept in Period 1, entered Period 2 and were randomized to receive Abatacept SC injections (fixed dose of 125 mg) starting on Day 85 and weekly for 12 weeks. Abatacept SC injections of 125 mg were continued in Reintroduction Period 3 and during the LTE Period until completion of the LTE.
- Placebo Received in Period 2: Participants who responded to abatacept in Period 1, entered Period 2 and were randomized to receive Placebo SC injections starting on Day 85 and weekly for 12 weeks. Abatacept SC injections of 125 mg were administered during Reintroduction Period 3 and during the LTE Period until completion of the LTE.
Arm/Group | Period 1 Non-Completers | Period 1 Non-Responders | Abatacept Received in Period 2 | Placebo Received in Period 2
Serious Adverse Events (participants affected / at risk) | 2/10 | 12/37 | 11/40 | 27/80
Other Adverse Events (participants affected / at risk) | 6/10 | 29/37 | 33/40 | 66/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 Non-Completers (N=10) | Period 1 Non-Responders (N=37) | Abatacept Received in Period 2 (N=40) | Placebo Received in Period 2 (N=80)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lupus nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 Non-Completers (N=10) | Period 1 Non-Responders (N=37) | Abatacept Received in Period 2 (N=40) | Placebo Received in Period 2 (N=80)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4
Folliculitis (Infections and infestations) | 0 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 3 | 2
Headache (Nervous system disorders) | 1 | 2 | 2 | 4
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Oedema peripheral (General disorders) | 1 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 2 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 3
Streptococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 3 | 3
Bronchitis (Infections and infestations) | 0 | 11 | 9 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 6
Depression (Psychiatric disorders) | 0 | 1 | 4 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 4
Herpes zoster (Infections and infestations) | 1 | 2 | 1 | 5
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 14 | 12 | 18
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 4
Gastroenteritis (Infections and infestations) | 0 | 3 | 1 | 6
Influenza (Infections and infestations) | 0 | 9 | 5 | 14
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Pharyngitis (Infections and infestations) | 0 | 3 | 3 | 7
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 5
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 3
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 5
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 2 | 6
Hypertension (Vascular disorders) | 0 | 3 | 3 | 10
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1 | 4
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2 | 3
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 5
Laryngitis (Infections and infestations) | 0 | 0 | 2 | 3
Sinusitis (Infections and infestations) | 1 | 6 | 6 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 3 | 7
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 6
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 4
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2
Animal bite (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 6 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 4
Localised infection (Infections and infestations) | 0 | 2 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Acute sinusitis (Infections and infestations) | 0 | 2 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 2 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Hepatic steatosis (Hepatobiliary disorders) | 0 | 2 | 0 | 3
Influenza like illness (General disorders) | 0 | 1 | 1 | 7
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 4
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 4 | 6 | 8
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 3
Urinary tract infection (Infections and infestations) | 0 | 6 | 10 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.